CLINICAL TRIAL: NCT03173560
Title: A Randomized, Open-Label (Formerly Double-Blind), Phase 2 Trial to Assess Safety and Efficacy of Lenvatinib at Two Different Starting Doses (18 mg vs. 14 mg QD) in Combination With Everolimus (5 mg QD) in Renal Cell Carcinoma Following One Prior VEGF-Targeted Treatment
Brief Title: Trial to Assess Safety and Efficacy of Lenvatinib (18 mg vs. 14 mg) in Combination With Everolimus in Participants With Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-218; 2016-002778-11 (EudraCT Number)
Record Dates: First submitted 2017-05-22; First posted 2017-06-02 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; lenvatinib; everolimus; E7080; VEGF-targeted treatment
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Masking Description: Study was initially double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib 14 mg plus everolimus 5 mg (Experimental): Participants will receive oral lenvatinib 14 mg once daily (QD) plus oral everolimus 5 mg QD as the starting dose for Cycle 1. If there are no intolerable Grade 2 or any >= Grade 3 treatment-emergent adverse events (TEAEs) that require dose reduction in the first 28-day cycle (that is, the first 4 weeks of treatment), the lenvatinib dose will be escalated to 18 mg QD (plus everolimus 5 mg) beginning in Cycle 2 or later (cycle length equal to [=] 28 days) during randomization phase. After the data cutoff for the primary analysis, participants will receive study treatment as continuous 56-day cycles.
  Interventions: Drug: lenvatinib; Drug: everolimus
- Lenvatinib 18 mg plus everolimus 5 mg (Experimental): Participants will receive oral lenvatinib 18 mg QD plus oral everolimus 5 mg QD as the starting dose in Cycle 1 or later (cycle length =28 days) during randomization phase. After the data cutoff for the primary analysis, participants will receive study treatment as continuous 56-day cycles.
  Interventions: Drug: lenvatinib; Drug: everolimus

INTERVENTIONS:
Drug: lenvatinib — lenvatinib capsules.
Drug: everolimus — everolimus tablets.

SUMMARY:
Study E7080-G000-218 is a Randomized, open-label (formerly Double-blind), Phase 2 Trial conducted to assess whether a starting dose of lenvatinib 14 milligrams (mg) in combination with everolimus 5 mg once daily (QD) will provide comparable efficacy (based on objective response rate [ORR] at 24 weeks [ORR24W]) with an improved safety profile compared to lenvatinib 18 mg in combination with everolimus 5 mg (based on treatment-emergent intolerable Grade 2, or any greater than or equal to (>=) Grade 3 adverse events (AEs) in the first 24 weeks after randomization).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of predominant clear cell renal cell carcinoma (RCC) (original tissue diagnosis of RCC is acceptable)
* Documented evidence of advanced RCC
* One prior disease progression episode on or after vascular endothelial growth factor (VEGF)-targeted treatment (for example, but not limited to, sunitinib, sorafenib, pazopanib, cabozantinib, bevacizumab, axitinib, vatalanib, AV951/tivozanib) administered for the treatment of RCC. Prior programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) treatment in addition to 1 prior VEGF-targeted treatment is allowed.
* At least 1 measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) meeting the following criteria:

  * Lymph node (LN) lesion that measures at least 1 dimension as >=1.5 centimeter (cm) in the short axis;
  * Non-nodal lesion that measures >=1.0 cm in the longest diameter;
  * The lesion is suitable for repeat measurement using computerized tomography/magnetic resonance imaging (CT/MRI). Lesions that have had external beam radiotherapy (EBRT) or locoregional therapy must show radiographic evidence of disease progression based on RECIST 1.1 to be deemed a target lesion.
* Male or female participants age >=18 years (or any age >=18 years if that age is considered to be an adult per the local jurisdiction) at the time of informed consent
* Karnofsky Performance Status (KPS) of >=70
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to (<=) 150/90 millimeters of mercury (mmHg) at Screening and no change in antihypertensive medications within 1 week before Cycle 1/Day 1
* Adequate renal function defined as calculated creatinine clearance >=30 milliliters per minute (mL/min) per the Cockcroft and Gault formula
* Adequate bone marrow function defined by:

  * Absolute neutrophil count (ANC) >=1500/millimeters cubed (mm^3) (>=1.5*10^9/Liters [L]);
  * Platelets >=100,000/mm^3 (>=100*10^9/L);
  * Hemoglobin >=9 grams per deciliter (g/dL)
* Adequate blood coagulation function defined by International Normalized Ratio (INR) <=1.5 (except for participants on warfarin therapy where INR must be <=3.0 prior to randomization)
* Adequate liver function defined by:

  * Total bilirubin <=1.5 times the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome;
  * Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3* the ULN (in the case of liver metastases <=5* the ULN). Participants with bone metastases with ALP values greater than 3 times can be included.
* Participant must voluntarily agree to provide written informed consent
* Participant must be willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* More than 1 prior VEGF-targeted treatment for advanced RCC
* Participants with Central Nervous System (CNS) metastases are not eligible, unless they have completed local therapy for at least 4 weeks and have discontinued the use of corticosteroids for this indication or are on a tapering regimen of corticosteroids (defined as <=10 mg prednisolone equivalent) before starting treatment in this study. Any signs (example, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
* Active malignancy (except for RCC or definitively treated basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or bladder) within the past 24 months
* Any anti-cancer treatment (except for radiation therapy) within 21 days, or any investigational agent within 30 days prior to the first dose of study drug; participants should have recovered from any toxicity related to previous anti-cancer treatment to Common Toxicity Criteria (CTC) grade 0 or 1.
* Prior radiation therapy within 21 days prior to the start of study treatment with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks prior to study treatment start
* Known intolerance to study drug (or any of the excipients) and/or known hypersensitivity to rapamycins (example, sirolimus, everolimus, temsirolimus) or any of the excipients
* Participants with proteinuria greater than (>) 1+ on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein >=1 g/24 hour will be ineligible.
* Fasting total cholesterol ˃300 mg/dL (or ˃7.75 millimoles [mmol]/L) and/or fasting triglycerides level ˃2.5* the ULN. Note: these participants can be included after initiation or adjustment of lipid-lowering medication.
* Uncontrolled diabetes as defined by fasting glucose >1.5 times the ULN. Note: these participants can be included after initiation or adjustment of glucose-lowering medication.
* Prolongation of QT corrected (QTc) interval to >480 milliseconds (ms)
* Participants who have not recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib or everolimus
* Bleeding or thrombotic disorders or participants at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (example, carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
* Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Significant cardiovascular impairment within 6 months prior to the first dose of study drug; history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke, or cardiac arrhythmia associated with significant cardiovascular impairment or left ventricular ejection fraction (LVEF) below the institutional normal range as determined by screening multigated acquisition (MUGA) scan or echocardiogram.
* Active infection (any infection requiring systemic treatment)
* Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of β-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Females of childbearing potential who (Note: all females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing].):

  * do not agree to use a highly effective method of contraception for the entire study period and for up to 8 weeks after study drug discontinuation, that is:

    * total abstinence (if it is their preferred and usual lifestyle)
    * an intrauterine device (IUD) or hormone releasing system (IUS)
    * a contraceptive implant
    * an oral contraceptive (with additional barrier method) (Note: Participants must be on a stable dose of the same oral hormonal contraceptive product for at least 4 weeks before dosing with study drug and for the duration of the study.) OR
  * do not have a vasectomized partner with confirmed azoospermia

For sites outside of the European Union, it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double barrier methods of contraception, such as condom plus diaphragm or cervical/vault cap with spermicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - Innovative Clinical Research Institute, LLC, Whittier, California
  - Baptist Health Medical Group Oncology, LLC - US Oncology, Miami, Florida
  - Optimal Research, Honolulu, Hawaii
  - Oklahoma Cancer Specialist and Research Institute , LLC, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology PA - US Oncology, Fort Worth, Texas
- Australia (5):
  - Macquarie University, Macquarie Park, New South Wales
  - Northern Cancer Institute, Saint Leonards, Saint Leonards, New South Wales
  - Adelaide Cancer Center, Kurralta Park, South Australia
  - Sunshine Hospital, Saint Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (7):
  - Alberta Health Service - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute- University of Toronto, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce, Prague
- Finland (4):
  - Helsingin Yliopistollinen Keskussairaala, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun Yliopistollinen Keskussairaala, Turku
  - Vaasan Keskussairaala, Vaasa
- Greece (6):
  - Alexandra Hospital, Athens
  - Metropolitan hospital, Athens
  - University General Hospital of Patras, Pátrai
  - Interbalkan Medical Center of Thessaloniki, Pylaia
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Italy (4):
  - IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Presidio Ospedaliero San Donato, Arezzo
  - AORN A Cardarelli, Napoli
  - Azienda Ospedaliera San Camillo Forlanini, Roma
- Netherlands (3):
  - Leids Universitair Medisch Centrum, Leiden
  - Hagaziekenhuis, The Hague
  - MC Haaglanden, The Hague
- Poland (8):
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Copernicus PL Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - NZOZ Vesalius, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Opolskie Centrum Onkologii, Opole
  - Mrukmed. Lekarz Beata Madej-Mruk i Partner. Spolka Partnerska, Rzeszów
  - MAGODENT Sp. z o.o. Szpital Elblaska, Warsaw
- Portugal (5):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Champalimaud Cancer Center, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
- Romania (4):
  - Medisprof SRL, Cluj-Napoca
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sfantul Nectarie, Craiova
  - Oncocenter Clinical Oncology, Timișoara
- Russia (8):
  - Altay Regional Oncology Center, Barnaul
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Central Clinical Hospital With Polyclinic of President Administration of RF, Moscow
  - Moscow City Oncology Hospital #62, Moscow
  - Moscow Scientific Research Oncology Institute P.A. Herzen, Moscow
  - Federal State Institution Medical Radiology Research Center, Obninsk
  - Clinical Oncology Dispensary, Omsk
  - Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Chonnam National University Hwasun Hospital, Jeonam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital - Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul Saint Mary's Hospital, Seoul
- Spain (13):
  - Hospital Universitario A Coruna, A Coruña
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clinica Universidad Navarra, Pamplona
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Hospital, Manchester
  - Mount Vernon Hospital, Northwood
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergerot C, Young Rha S, Pal S, Koralewski P, Stroyakovskiy D, Alekseev B, Parnis F, Castellano D, Lyun Lee J, Sunela K, Ciuleanu T, Heng D, Glen H, Wang J, Bennett L, Pan J, O'Hara K, Puente J. Health-Related Quality of Life Outcomes With Two Different Starting Doses of Lenvatinib in Combination With Everolimus for Previously Treated Renal Cell Carcinoma. Oncologist. 2023 Jan 18;28(1):59-71. doi: 10.1093/oncolo/oyac142. PMID 35881028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 82 investigative sites in Australia, Korea, Taiwan, Czech, Poland, Romania, Russia, Finland, Greece, Italy, Netherlands, Portugal, Spain, United Kingdom, Canada and the United States from 17 August 2017 to 20 June 2024.
Pre-assignment Details: A total of 489 participants were screened, of which 146 were screen failures and 343 were enrolled and randomized, out of which 341 participants were treated.
Groups:
- Lenvatinib 14 mg + Everolimus 5 mg: Participants received lenvatinib 14 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily as the starting dose in a 28-day treatment cycle until progressive disease (PD), development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first. Participants who had no intolerable Grade 2 or any greater than or equal to (>=) Grade 3 treatment-emergent adverse events (TEAEs) that required dose reduction in the first 28-day cycle (that is, the first 4 weeks of treatment), had lenvatinib dose titrated to 18 mg once daily (along with everolimus 5 mg) beginning in Cycle 2 or later (cycle length equals to (=) 28 days) during randomization phase.
- Lenvatinib 18 mg + Everolimus 5 mg: Participants received lenvatinib 18 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily as the starting dose in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first.
Period: Overall Study
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Started | 172 | 171
Treated Participants | 172 | 169
Safety Set (One participant was randomized to lenvatinib 18 mg arm but received lenvatinib 14 mg as the starting dose and therefore was included in lenvatinib 14 mg arm in safety population.) | 173 | 168
Completed | 91 | 101
Not Completed | 81 | 70
Not completed — Death | 70 | 60
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Lenvatinib 14 mg + Everolimus 5 mg: Participants received lenvatinib 14 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily as the starting dose in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first. Participants who had no intolerable Grade 2 or any >=Grade 3 TEAEs that required dose reduction in the first 28-day cycle (that is, the first 4 weeks of treatment), had lenvatinib dose titrated to 18 mg once daily (along with everolimus 5 mg) beginning in Cycle 2 or later (cycle length =28 days) during randomization phase.
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg | Total
Number analyzed (Participants) | 172 | 171 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.59) | 61.5 (9.90) | 61.0 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 81
  Male | 133 | 129 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 168 | 163 | 331
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 27 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 137 | 140 | 277
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate at Week 24 (ORR24W)
Description: ORR24W was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) at the Week 24 (after randomization) time point, during treatment or within 28 days after the last dose date but on or prior to the start of new anticancer therapy based on investigator assessment according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 millimeters (mm). PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. To be considered a BOR, all responses had to be confirmed no less than 4 weeks after the initial assessment of response.
Time Frame: At Week 24
Population: Per-protocol analysis set 1 (PPAS1) included all randomized participants minus the 32 participants who had received >=2 incorrect lenvatinib doses due to interactive voice and web response system (IxRS) issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 156 | 155
percentage of participants | 32.1 [24.7 to 39.4] | 34.8 [27.3 to 42.3]
Statistical Analysis 1: Comparison: Lenvatinib 14 mg + Everolimus 5 mg vs Lenvatinib 18 mg + Everolimus 5 mg; Test type: Non-Inferiority — Odd ratio for ORR24W was analyzed along with 90% CI for each treatment arm using Cochran-Mantel-Haenszel (CMH) method, stratified by Memorial Sloan-Kettering Cancer Center (MSKCC) prognostic group and prior programmed cell death protein 1/ programmed cell death protein ligand 1 (PD-1/PD-L1) treatment from IxRS data. Non-inferiority would be claimed if 1-sided P value is <=0.045 at the final analysis for the non-inferiority test with the non-inferiority margin of the odd ratio =0.76; p = 0.2676, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 90% CI 2-sided [0.59 to 1.32]

2. Primary Outcome: Percentage of Participants With Intolerable Grade 2 or Any Grade >=Grade 3 TEAEs Within 24 Weeks
Description: TEAE was defined as an adverse event (AE) with an onset that had occurred after receiving study drug. A severity grade was defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. As per NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: Up to Week 24
Population: Per-protocol safety analysis set included all randomized and treated participants minus 32 participants who had received >=2 incorrect lenvatinib doses due to IxRS issues according to actual treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 157 | 152
percentage of participants | 82.8 [76.9 to 88.7] | 79.6 [73.2 to 86.0]
Statistical Analysis 1: Comparison: Lenvatinib 14 mg + Everolimus 5 mg vs Lenvatinib 18 mg + Everolimus 5 mg; Test type: Superiority — Percentage of participants with intolerable Grade 2 or any Grade >=Grade 3 TEAEs within 24 weeks was tested using CMH method at 2-sided α=0.05, stratified by MSKCC prognostic group and prior PD-1/PD-L1 treatment from IxRS data. The treatment difference and 95% CI were also calculated based on asymptotic normal approximation; p = 0.4763, Cochran-Mantel-Haenszel; Difference = 3.2, 95% CI 2-sided [-5.5 to 11.9]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of PD by investigator assessment or date of death, whichever occurred first according to RECIST v1.1. PD: at least 20% increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter (SOD) of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. Median PFS was analyzed using the Kaplan-Meier product-limit estimates for each treatment group and presented with 2-sided 95% confidence interval (CI). As pre-specified in the protocol, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: From the date of randomization to the date of the first documentation of PD or date of death, whichever occurred first or up to date of data cutoff for the primary analysis (up to 29 months)
Population: PPAS1 included all randomized participants minus the 32 participants who had received >=2 incorrect lenvatinib doses due to IxRS issues.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 156 | 155
months | 11.1 [9.0 to 12.9] | 14.7 [11.1 to 20.3]
Statistical Analysis 1: Comparison: Lenvatinib 14 mg + Everolimus 5 mg vs Lenvatinib 18 mg + Everolimus 5 mg; Test type: Other — The hazard ratio and the corresponding 90% CIs were estimated using the Cox regression model with Efron's method for ties, stratified by MSKCC prognostic group and prior PD-1/PD-L1 treatment; Hazard Ratio (HR) = 1.42, 90% CI 2-sided [1.08 to 1.86]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a BOR of CR or PR at the at the end of treatment based on investigator assessment according to RECIST v1.1. CR: defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR: defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. To be considered a BOR, all responses had to be confirmed no less than 4 weeks after the initial assessment of response. As pre-specified in the protocol, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: From date of randomization up to first documentation of PD or date of death, whichever occurred first or up to the date of data cut off for the primary analysis (up to 29 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 156 | 155
percentage of participants | 34.6 [27.1 to 42.1] | 40.6 [32.9 to 48.4]
Statistical Analysis 1: Comparison: Lenvatinib 14 mg + Everolimus 5 mg vs Lenvatinib 18 mg + Everolimus 5 mg; Test type: Other — Odd ratio for ORR was analyzed along with 90% CI for each treatment arm using CMH method stratified by MSKCC prognostic group and PD-1/PD-L1 treatment from IxRS data; Odds Ratio (OR) = 0.77, 90% CI 2-sided [0.52 to 1.14]

5. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs
Description: TEAEs were defined as those adverse events (AEs) that occurred (or worsened, if present at Baseline) after the first dose of study drug through 28 days after the last dose of study drug. An AE was defined as any untoward medical occurrence in a participants or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. A serious adverse event (SAE) was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: From date of first dose of study drug up to 28 days after last dose of study drug (up to 71 months)
Population: Safety analysis set (SAS) included all participants who were randomized and received at least 1 dose of study drug according to the treatment starting dose actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 173 | 168
Participants
  Participants With TEAEs | 173 | 167
  Participants With Serious TEAEs | 92 | 87

6. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Toxicity
Description: Percentage of participants who discontinued treatment due to toxicity, defined as the percentage of participants who discontinued study treatment due to TEAEs. Toxicity (except hypertension and non-infectious pneumonitis) was assessed according to NCI-CTCAE v4.03.
Time Frame: From date of first dose of study drug up to 28 days after last dose of study drug (up to 71 months)
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 172 | 171
percentage of participants | 17.4 | 25.1

7. Secondary Outcome: Time to Treatment Failure Due to Toxicity
Description: Time to treatment failure due to toxicity was defined as the time from the date of randomization to the date that a participant discontinued study treatment due to TEAEs. Toxicity (except hypertension and non-infectious pneumonitis) was assessed according to CTCAE v4.03. As planned, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: From the date of randomization to the date of discontinuation of study treatment due to TEAEs, or date of data cut off for the primary analysis (up to 29 months)
Population: FAS included all randomized participants.
Measure: Median (Full Range); unit: months
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 172 | 171
months | 3.15 [0.5 to 12.7] | 5.70 [0.8 to 24.6]

8. Secondary Outcome: Plasma Concentration of Lenvatinib
Description: PK sparse sampling was performed. As planned, the post-dose plasma sample was collected anytime between 0.5 to 4 hours at Cycle 1 Days 1 and 15, between 6 to 10 hours at Cycle 1 Days 1 and 15, and between 2 to 12 hours at Cycle 2 Day 1. Only one sample was collected for each post-dose category between specified timepoints.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours post-dose; Cycle 1 Day 15: pre-dose, 0.5-4 hours and 6-10 hours post-dose; Cycle 2 Day 1: pre-dose and 2-12 hours post-dose (each cycle length =28 days)
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug with documented dosing history and had at least 1 evaluable lenvatinib plasma or everolimus whole blood concentration data. Here, "overall number of participants analyzed" are the participants who were evaluable for the outcome measure and "number analyzed" were the participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 168 | 160
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: 0.5-4 hours post-dose | 57.9 (96.54) | 82.3 (119.89)
  Cycle 1 Day 1: 6-10 hours post-dose: number analyzed (Participants) | 166 | 154
  Cycle 1 Day 1: 6-10 hours post-dose | 136.3 (66.53) | 193.7 (93.08)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 154 | 149
  Cycle 1 Day 15: Pre-dose | 53.7 (62.31) | 64.0 (59.71)
  Cycle 1 Day 15: 0.5-4 hours post-dose: number analyzed (Participants) | 147 | 147
  Cycle 1 Day 15: 0.5-4 hours post-dose | 99.6 (102.54) | 133.4 (125.65)
  Cycle 1 Day 15: 6-10 hours post-dose: number analyzed (Participants) | 148 | 143
  Cycle 1 Day 15: 6-10 hours post-dose | 177.8 (89.42) | 236.2 (135.21)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 160 | 151
  Cycle 2 Day 1: Pre-dose | 42.8 (42.84) | 50.6 (46.06)
  Cycle 2 Day 1: 2-12 hours post-dose: number analyzed (Participants) | 154 | 143
  Cycle 2 Day 1: 2-12 hours post-dose | 172.8 (130.90) | 190.3 (114.85)

9. Secondary Outcome: Whole Blood Concentration of Everolimus
Description: PK sparse sampling was performed. As planned, the post-dose whole blood sample was collected anytime between 0.5 to 4 hours at Cycle 1 Days 1 and 15, between 6 to 10 hours at Cycle 1 Days 1 and 15, and between 2 to 12 hours at Cycle 2 Day 1. Only one sample was collected for each post-dose category between specified timepoints.
Time Frame: as for outcome 8
Population: PK analysis set included all participants who received at least 1 dose of study drug with documented dosing history and had at least 1 evaluable lenvatinib plasma or everolimus whole blood concentration data. Here, "overall number of participants analyzed" are the participants who were evaluable for the outcome measure and "number analyzed" were the participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 120 | 117
ng/mL
  Cycle 1 Day 1: 0.5-4 hours post-dose: number analyzed (Participants) | 106 | 117
  Cycle 1 Day 1: 0.5-4 hours post-dose | 18.3 (15.89) | 18.6 (16.39)
  Cycle 1 Day 1: 6-10 hours post-dose: number analyzed (Participants) | 103 | 115
  Cycle 1 Day 1: 6-10 hours post-dose | 9.2 (6.60) | 8.4 (5.64)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 110 | 111
  Cycle 1 Day 15: Pre-dose | 8.4 (4.84) | 7.4 (5.51)
  Cycle 1 Day 15: 0.5-4 hours post-dose: number analyzed (Participants) | 106 | 111
  Cycle 1 Day 15: 0.5-4 hours post-dose | 23.7 (15.41) | 23.4 (16.96)
  Cycle 1 Day 15: 6-10 hours post-dose: number analyzed (Participants) | 107 | 106
  Cycle 1 Day 15: 6-10 hours post-dose | 14.3 (5.83) | 14.3 (9.22)
  Cycle 2 Day 1: Pre-dose | 7.8 (5.44) | 5.9 (4.02)
  Cycle 2 Day 1: 2-12 hours post-dose: number analyzed (Participants) | 112 | 112
  Cycle 2 Day 1: 2-12 hours post-dose | 22.9 (12.67) | 19.5 (9.74)

10. Secondary Outcome: Model Predicted Apparent Total Clearance (CL/F) for Lenvatinib Alone and When Coadministration With Everolimus in Renal Cell Carcinoma (RCC) Participants to Assess Drug-Drug Interaction
Description: Sparse PK samples were collected and analyzed using a population PK approach to estimate PK parameters. The lenvatinib concentration data was pooled from studies E7080 -G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) and from current study E7080-G000-218 (NCT03173560). A previously developed 3-compartment PK model for lenvatinib was fitted to the pooled dataset. Individual lenvatinib CL/F value was derived from the final PK model. The outcome measure was assessed for lenvatinib 18 mg dose only.
Time Frame: as for outcome 8
Population: PK analysis set included all participants who received at least 1 dose of study drug with documented dosing history and had at least 1 evaluable lenvatinib plasma concentration data. Population included participants from E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) and current study E7080-G000-218 (NCT03173560). Here, "overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Groups:
- Lenvatinib 18 mg: Participants with RCC received lenvatinib 18 mg, capsule, orally, once daily until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up or until the end of the study, whichever occurred first in studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) and in this current study E7080-G000-218 (NCT03173560).
- Lenvatinib 18 mg + Everolimus 5 mg: Participants with RCC received lenvatinib 18 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up or until the end of the study, whichever occurred first in studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) and in this current study E7080-G000-218 (NCT03173560).
Arm/Group | Lenvatinib 18 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 48 | 443
liter per hour (L/h) | 6.37 (2.01) | 5.77 (2.01)

11. Secondary Outcome: Model Predicted Dose Normalized Area Under the Plasma Concentration-time Curve (AUC) for Lenvatinib Alone and When Coadministration With Everolimus in RCC Participants to Assess Drug-Drug Interaction
Description: Sparse PK samples were collected and analyzed using a population PK approach to estimate PK parameters. The lenvatinib concentration data was pooled from studies E7080 -G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) and from current study E7080-G000-218 (NCT03173560). A previously developed 3-compartment PK model for lenvatinib was fitted to the pooled dataset. Individual lenvatinib AUC at steady state based on the starting dose was derived as a function of starting dose from the final PK model. The outcome measure was assessed for lenvatinib 18 mg dose only.
Time Frame: as for outcome 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lenvatinib 18 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 48 | 443
nanogram*hour per milliliter (ng*h/mL) | 3693 (1295) | 4350 (2934)

12. Secondary Outcome: Model Predicted CL/F for Everolimus Alone and When Coadministration With Lenvatinib in RCC Participants to Assess Drug-Drug Interaction
Description: Sparse PK samples were collected and analyzed using a population PK approach to estimate PK parameters. The everolimus concentration data was pooled from studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) or from current study E7080-G000-218 (NCT03173560). A previously developed 3-compartment PK model for everolimus was fitted to the pooled dataset. Individual everolimus CL/F value was derived from the final PK model.
Time Frame: as for outcome 8
Population: PK analysis set included all participants who received at least 1 dose of study drug with documented dosing history and had at least 1 evaluable everolimus whole blood concentration data. Population included participants from E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) or current study E7080-G000-218 (NCT03173560). Here, "overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Groups:
- Everolimus 10 mg: Participants with RCC received everolimus 10 mg, capsule, orally, once daily until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up or until the end of the study, whichever occurred first in studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) or in this current study E7080-G000-218 (NCT03173560).
- Lenvatinib + Everolimus 5 mg: Participants with RCC received lenvatinib 12 to 24 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up or until the end of the study, whichever occurred first in studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) or in this current study E7080-G000-218 (NCT03173560).
Arm/Group | Everolimus 10 mg | Lenvatinib + Everolimus 5 mg
Number analyzed (Participants) | 33 | 345
liter per hour (L/h) | 22.3 (10.5) | 19.4 (7.9)

13. Secondary Outcome: Model Predicted Dose Normalized AUC for Everolimus Alone and When Coadministration With Lenvatinib in RCC Participants to Assess Drug-Drug Interaction
Description: Sparse PK samples were collected and analyzed using a population PK approach to estimate PK parameters. The everolimus concentration data was pooled from studies E7080-G000-205 (NCT01136733), E7080-M001-221 (NCT02915783), E7080-J081-112 (NCT02454478) or from current study E7080-G000-218 (NCT03173560). A previously developed 3-compartment PK model for everolimus was fitted to the pooled dataset. Individual everolimus AUC at steady state based on the starting dose was derived as a function of starting dose from the final PK model.
Time Frame: as for outcome 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Everolimus 10 mg | Lenvatinib + Everolimus 5 mg
Number analyzed (Participants) | 33 | 345
ng*hour/mL | 507.4 (176.6) | 305.5 (174.0)

14. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. In the absence of confirmation of death, participants will be censored either at the date that the participant was last known to be alive or the date of data cutoff for the primary analysis, whichever comes earlier. Median OS was to be calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval. As pre-specified in the protocol, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: From the date of randomization until the date of death from any cause, or up to date of data cut off for the primary analysis (up to 29 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 156 | 155
months | 27.0 [18.3 to NA] — Upper limit of 95% CI was not estimable because insufficient number of participants had events. | NA [23.8 to NA] — Median and upper limit of 95% CI was not estimable because insufficient number of participants had events.

15. Secondary Outcome: Health-Related Quality of Life (HRQoL) Assessed by Functional Assessment of Cancer Therapy Kidney Syndrome Index-Disease-Related Symptoms (FKSI-DRS) Scores
Description: The FKSI-DRS consisted of 9 items that experts and participants had indicated are important targets for the treatment of advanced kidney cancer, and that clinical experts had indicated are primarily disease-related, as opposed to treatment-related. Symptoms assessed on the FKSI-DRS included lack of energy, fatigue, weight loss, pain, bone pain, shortness of breath, cough, fever, or hematuria. Each item was scored on a 5-point Likert-type scale (0 = not at all; 4 = very much) where total score ranged from 0 (worst) to 36 (best), where higher scores correspond to better outcomes. As pre-specified in the protocol, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: At baseline (prior to first dose of study drug), on Day 1 of each subsequent cycle (cycle length =28 days), and at the Off-treatment visit (up to 29 months)
Population: Quality of Life (QoL) analysis set consisted of all participants who had any QoL data. Here "overall number of participants analyzed" are the participants who were evaluable for the outcome measure and "number analyzed" were the participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 169 | 162
score on a scale
  Baseline | 29.69 (4.819) | 29 (5.886)
  Cycle 2 Day 1: number analyzed (Participants) | 156 | 152
  Cycle 2 Day 1 | 28.43 (5.269) | 28.31 (5.162)
  Cycle 3 Day 1: number analyzed (Participants) | 146 | 140
  Cycle 3 Day 1 | 28.26 (5.344) | 28.80 (5.455)
  Cycle 4 Day 1: number analyzed (Participants) | 133 | 137
  Cycle 4 Day 1 | 27.97 (5.524) | 29.11 (5.183)
  Cycle 5 Day 1: number analyzed (Participants) | 125 | 127
  Cycle 5 Day 1 | 28 (5.680) | 29.14 (5.081)
  Cycle 6 Day 1: number analyzed (Participants) | 120 | 120
  Cycle 6 Day 1 | 28.63 (5.185) | 29.46 (5.107)
  Cycle 7 Day 1: number analyzed (Participants) | 105 | 103
  Cycle 7 Day 1 | 28.31 (5.486) | 29.58 (4.803)
  Cycle 8 Day 1: number analyzed (Participants) | 96 | 97
  Cycle 8 Day 1 | 28.36 (6.204) | 29.85 (4.610)
  Cycle 9 Day 1: number analyzed (Participants) | 89 | 92
  Cycle 9 Day 1 | 28.58 (5.562) | 29.84 (5.005)
  Cycle 10 Day 1: number analyzed (Participants) | 79 | 75
  Cycle 10 Day 1 | 29.10 (5.294) | 30.70 (4.297)
  Cycle 11 Day 1: number analyzed (Participants) | 68 | 72
  Cycle 11 Day 1 | 29.56 (5.035) | 30.09 (5.316)
  Cycle 12 Day 1: number analyzed (Participants) | 64 | 61
  Cycle 12 Day 1 | 29.34 (5.149) | 30.75 (5.127)
  Cycle 13 Day 1: number analyzed (Participants) | 56 | 53
  Cycle 13 Day 1 | 29.26 (4.851) | 30.93 (4.201)
  Cycle 14 Day 1: number analyzed (Participants) | 48 | 52
  Cycle 14 Day 1 | 29.81 (4.752) | 31.06 (4.830)
  Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Cycle 15 Day 1 | 30.09 (5.121) | 30.52 (4.417)
  Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Cycle 16 Day 1 | 29.93 (5.293) | 30.91 (4.704)
  Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Cycle 17 Day 1 | 29.36 (5.233) | 31.52 (4.875)
  Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Cycle 18 Day 1 | 29.81 (4.293) | 31.41 (4.639)
  Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Cycle 19 Day 1 | 28.48 (6.216) | 30.82 (4.469)
  Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Cycle 20 Day 1 | 28.77 (6.058) | 30.69 (4.575)
  Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Cycle 21 Day 1 | 29.35 (4.707) | 32 (3.243)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Cycle 22 Day 1 | 30.32 (4.978) | 30.59 (5.168)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Cycle 23 Day 1 | 30.53 (3.998) | 30.29 (5.544)
  Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Cycle 24 Day 1 | 29.47 (5.041) | 31.58 (3.977)
  Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Cycle 25 Day 1 | 27.92 (6.388) | 31.69 (4.270)
  Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Cycle 26 Day 1 | 28.75 (4.862) | 29.82 (6.422)
  Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Cycle 27 Day 1 | 29.83 (5.345) | 32.86 (2.854)
  Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 28 Day 1 | 30.50 (4.435) | 33.67 (1.862)
  Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Cycle 29 Day 1 | 29.50 (4.359) | 33.40 (1.342)
  Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Cycle 30 Day 1 | 30.75 (4.031) | 36
  Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 31 Day 1 | 31 |
  Off-treatment Visit: number analyzed (Participants) | 78 | 74
  Off-treatment Visit | 27.42 (5.953) | 27.86 (6.500)

16. Secondary Outcome: HRQoL Assessed by European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 Scores
Description: The EORT QLQ-C30 consisted of 30 questions comprising 9 multiple-item scales and 6 single items. Multiple-item scales of QLQ-C30 consisted of 5 functional scales (physical, role, emotional, cognitive, and social) and 3 symptom scales (fatigue, nausea and vomiting, pain) and a global health status/QOL score. Six single-item scales of QLQ-C30 involved dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. First 28 questions used a 4-point scale (1 = Not at all to 4 = Very much); and last 2 questions used a 7-point scale (1 = Very poor to 7 = Excellent). Scores for all scales range from 0 to 100. For the overall HRQoL and functioning scales, a higher score was correlated with better HRQoL, whereas a higher score for symptom scales represented worse HRQoL. As pre-specified in protocol, data for secondary outcome measure was collected and analyzed till primary analysis only.
Time Frame: as for outcome 15
Population: QoL analysis set consisted of all participants who had any QoL data. Here, overall number of participants analyzed" are the participants who were evaluable for the outcome measure and "number analyzed" were the participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 171 | 162
score on a scale
  Global Health Status/QoL Score; Baseline | 63.35 (22.020) | 63.58 (21.340)
  Global Health Status/QoL Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 151
  Global Health Status/QoL Score; Cycle 2 Day 1 | 58.60 (21.234) | 60.93 (20.280)
  Global Health Status/QoL Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 142
  Global Health Status/QoL Score; Cycle 3 Day 1 | 56.43 (24.065) | 61.85 (20.202)
  Global Health Status/QoL Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 136
  Global Health Status/QoL Score; Cycle 4 Day 1 | 58.71 (19.754) | 62.62 (19.641)
  Global Health Status/QoL Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 126
  Global Health Status/QoL Score; Cycle 5 Day 1 | 59.38 (21.670) | 63.76 (20.339)
  Global Health Status/QoL Score; Cycle 6 Day 1: number analyzed (Participants) | 120 | 119
  Global Health Status/QoL Score; Cycle 6 Day 1 | 58.75 (21.028) | 63.73 (19.756)
  Global Health Status/QoL Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Global Health Status/QoL Score; Cycle 7 Day 1 | 58.72 (20.134) | 62.54 (20.153)
  Global Health Status/QoL Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Global Health Status/QoL Score; Cycle 8 Day 1 | 58.68 (20.409) | 62.11 (20.271)
  Global Health Status/QoL Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Global Health Status/QoL Score; Cycle 9 Day 1 | 58.97 (18.726) | 63.77 (20.429)
  Global Health Status/QoL Score; Cycle 10 Day 1: number analyzed (Participants) | 80 | 74
  Global Health Status/QoL Score; Cycle 10 Day 1 | 63.13 (19.612) | 66.44 (19.012)
  Global Health Status/QoL Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Global Health Status/QoL Score; Cycle 11 Day 1 | 60.87 (18.705) | 65.86 (21.173)
  Global Health Status/QoL Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 60
  Global Health Status/QoL Score; Cycle 12 Day 1 | 57.81 (18.891) | 66.94 (18.409)
  Global Health Status/QoL Score; Cycle 13 Day 1: number analyzed (Participants) | 55 | 55
  Global Health Status/QoL Score; Cycle 13 Day 1 | 59.39 (19.047) | 68.94 (18.388)
  Global Health Status/QoL Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Global Health Status/QoL Score; Cycle 14 Day 1 | 61.56 (17.498) | 70.35 (15.605)
  Global Health Status/QoL Score; Cycle 15 Day 1: number analyzed (Participants) | 43 | 51
  Global Health Status/QoL Score; Cycle 15 Day 1 | 62.98 (16.795) | 66.83 (16.955)
  Global Health Status/QoL Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Global Health Status/QoL Score; Cycle 16 Day 1 | 61.59 (17.567) | 64.54 (19.386)
  Global Health Status/QoL Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Global Health Status/QoL Score; Cycle 17 Day 1 | 60.88 (16.882) | 67.71 (18.794)
  Global Health Status/QoL Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Global Health Status/QoL Score; Cycle 18 Day 1 | 59.68 (16.258) | 68.38 (17.859)
  Global Health Status/QoL Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Global Health Status/QoL Score; Cycle 19 Day 1 | 58.33 (19.747) | 66.67 (15.215)
  Global Health Status/QoL Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Global Health Status/QoL Score; Cycle 20 Day 1 | 58.95 (18.479) | 66.40 (15.736)
  Global Health Status/QoL Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Global Health Status/QoL Score; Cycle 21 Day 1 | 57.05 (18.362) | 71.13 (15.463)
  Global Health Status/QoL Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Global Health Status/QoL Score; Cycle 22 Day 1 | 62.72 (14.532) | 66.05 (17.438)
  Global Health Status/QoL Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Global Health Status/QoL Score; Cycle 23 Day 1 | 60 (15.494) | 66.67 (14.948)
  Global Health Status/QoL Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Global Health Status/QoL Score; Cycle 24 Day 1 | 64.44 (17.385) | 65.79 (18.818)
  Global Health Status/QoL Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Global Health Status/QoL Score; Cycle 25 Day 1 | 58.33 (16.667) | 69.79 (14.868)
  Global Health Status/QoL Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Global Health Status/QoL Score; Cycle 26 Day 1 | 59.38 (15.064) | 60.90 (18.442)
  Global Health Status/QoL Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Global Health Status/QoL Score; Cycle 27 Day 1 | 59.72 (18.572) | 71.43 (18.545)
  Global Health Status/QoL Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Global Health Status/QoL Score; Cycle 28 Day 1 | 58.33 (21.517) | 77.78 (13.608)
  Global Health Status/QoL Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Global Health Status/QoL Score; Cycle 29 Day 1 | 56.25 (18.478) | 75 (16.667)
  Global Health Status/QoL Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Global Health Status/QoL Score; Cycle 30 Day 1 | 54.17 (15.957) | 66.67
  Global Health Status/QoL Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Global Health Status/QoL Score; Cycle 31 Day 1 | 33.33 |
  Global Health Status/QoL Score; Off-treatment Visit: number analyzed (Participants) | 80 | 73
  Global Health Status/QoL Score; Off-treatment Visit | 51.04 (23.133) | 56.05 (22.363)
  Physical Functioning Score; Baseline | 76.36 (19.282) | 76.60 (21.855)
  Physical Functioning Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 150
  Physical Functioning Score; Cycle 2 Day 1 | 73.54 (19.857) | 75.38 (19.706)
  Physical Functioning Score; Cycle 3 Day 1: number analyzed (Participants) | 148 | 142
  Physical Functioning Score; Cycle 3 Day 1 | 72.74 (21.227) | 76.15 (19.160)
  Physical Functioning Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 137
  Physical Functioning Score; Cycle 4 Day 1 | 70.90 (20.873) | 75.40 (20.155)
  Physical Functioning Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 127
  Physical Functioning Score; Cycle 5 Day 1 | 72.80 (19.284) | 77.85 (18.342)
  Physical Functioning Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Physical Functioning Score; Cycle 6 Day 1 | 72.17 (21.694) | 77.76 (18.562)
  Physical Functioning Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Physical Functioning Score; Cycle 7 Day 1 | 73.02 (20.769) | 78.41 (18.034)
  Physical Functioning Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Physical Functioning Score; Cycle 8 Day 1 | 72.77 (20.422) | 79.11 (17.707)
  Physical Functioning Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Physical Functioning Score; Cycle 9 Day 1 | 74.54 (19.389) | 80.60 (16.041)
  Physical Functioning Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Physical Functioning Score; Cycle 10 Day 1 | 75.06 (18.908) | 81.20 (16.271)
  Physical Functioning Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Physical Functioning Score; Cycle 11 Day 1 | 73.72 (18.073) | 81.13 (16.638)
  Physical Functioning Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Physical Functioning Score; Cycle 12 Day 1 | 75.52 (17.080) | 83.01 (15.254)
  Physical Functioning Score; Cycle 13 Day 1: number analyzed (Participants) | 55 | 55
  Physical Functioning Score; Cycle 13 Day 1 | 74.55 (17.874) | 80.24 (16.873)
  Physical Functioning Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Physical Functioning Score; Cycle 14 Day 1 | 75.78 (16.925) | 82.39 (16.387)
  Physical Functioning Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Physical Functioning Score; Cycle 15 Day 1 | 75.45 (16.629) | 80.92 (17.283)
  Physical Functioning Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Physical Functioning Score; Cycle 16 Day 1 | 73.46 (17.129) | 81.74 (15.982)
  Physical Functioning Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Physical Functioning Score; Cycle 17 Day 1 | 71.85 (17.896) | 82.33 (15.657)
  Physical Functioning Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Physical Functioning Score; Cycle 18 Day 1 | 75.48 (17.838) | 81.52 (16.135)
  Physical Functioning Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Physical Functioning Score; Cycle 19 Day 1 | 76.67 (15.771) | 81.57 (16.002)
  Physical Functioning Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Physical Functioning Score; Cycle 20 Day 1 | 73.09 (22.071) | 82.80 (13.854)
  Physical Functioning Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Physical Functioning Score; Cycle 21 Day 1 | 74.62 (18.668) | 84.29 (12.335)
  Physical Functioning Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Physical Functioning Score; Cycle 22 Day 1 | 80.35 (14.483) | 82.72 (15.164)
  Physical Functioning Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Physical Functioning Score; Cycle 23 Day 1 | 79.56 (14.357) | 81.39 (17.248)
  Physical Functioning Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Physical Functioning Score; Cycle 24 Day 1 | 77.33 (16.676) | 83.86 (13.755)
  Physical Functioning Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Physical Functioning Score; Cycle 25 Day 1 | 72.78 (15.688) | 84.17 (15.753)
  Physical Functioning Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Physical Functioning Score; Cycle 26 Day 1 | 76.67 (6.172) | 71.79 (29.833)
  Physical Functioning Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Physical Functioning Score; Cycle 27 Day 1 | 76.67 (6.992) | 85.71 (16.523)
  Physical Functioning Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Physical Functioning Score; Cycle 28 Day 1 | 78.33 (3.333) | 90 (15.635)
  Physical Functioning Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Physical Functioning Score; Cycle 29 Day 1 | 78.33 (3.333) | 86.67 (16.330)
  Physical Functioning Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Physical Functioning Score; Cycle 30 Day 1 | 76.67 (3.849) | 100
  Physical Functioning Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Physical Functioning Score; Cycle 31 Day 1 | 80 |
  Physical Functioning Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Physical Functioning Score; Off-treatment Visit | 64.50 (25.891) | 70.41 (25.139)
  Role Functioning Score; Baseline | 73.78 (27.471) | 75.72 (27.932)
  Role Functioning Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 150
  Role Functioning Score; Cycle 2 Day 1 | 68.25 (27.951) | 69.33 (27.449)
  Role Functioning Score; Cycle 3 Day 1: number analyzed (Participants) | 148 | 142
  Role Functioning Score; Cycle 3 Day 1 | 67 (28.136) | 72.18 (25.630)
  Role Functioning Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 137
  Role Functioning Score; Cycle 4 Day 1 | 66.67 (27.993) | 73.60 (26.169)
  Role Functioning Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 127
  Role Functioning Score; Cycle 5 Day 1 | 67.32 (28.479) | 72.44 (25.143)
  Role Functioning Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Role Functioning Score; Cycle 6 Day 1 | 68.16 (27.245) | 73.75 (27.557)
  Role Functioning Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Role Functioning Score; Cycle 7 Day 1 | 66.51 (27.424) | 73.97 (25.205)
  Role Functioning Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Role Functioning Score; Cycle 8 Day 1 | 68.20 (27.712) | 75.60 (26.139)
  Role Functioning Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Role Functioning Score; Cycle 9 Day 1 | 67.58 (26.101) | 75.91 (25.242)
  Role Functioning Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Role Functioning Score; Cycle 10 Day 1 | 68.52 (27.131) | 76.89 (24.027)
  Role Functioning Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Role Functioning Score; Cycle 11 Day 1 | 69.57 (25.237) | 79.11 (23.691)
  Role Functioning Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Role Functioning Score; Cycle 12 Day 1 | 70.51 (24.785) | 80.91 (22.953)
  Role Functioning Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Role Functioning Score; Cycle 13 Day 1 | 69.64 (24.434) | 80 (24.721)
  Role Functioning Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Role Functioning Score; Cycle 14 Day 1 | 71.09 (24.242) | 81.13 (23.121)
  Role Functioning Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Role Functioning Score; Cycle 15 Day 1 | 72.73 (22.184) | 74.84 (25.685)
  Role Functioning Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Role Functioning Score; Cycle 16 Day 1 | 70.33 (23.426) | 79.08 (21.272)
  Role Functioning Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Role Functioning Score; Cycle 17 Day 1 | 65.74 (22.868) | 83.75 (18.292)
  Role Functioning Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Role Functioning Score; Cycle 18 Day 1 | 67.74 (20.609) | 82.35 (22.073)
  Role Functioning Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Role Functioning Score; Cycle 19 Day 1 | 67.28 (28.300) | 77.45 (23.883)
  Role Functioning Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Role Functioning Score; Cycle 20 Day 1 | 70.37 (23.266) | 79.57 (24.612)
  Role Functioning Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Role Functioning Score; Cycle 21 Day 1 | 69.23 (21.956) | 81.55 (19.948)
  Role Functioning Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Role Functioning Score; Cycle 22 Day 1 | 75.44 (20.313) | 77.78 (22.169)
  Role Functioning Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Role Functioning Score; Cycle 23 Day 1 | 73.33 (25.040) | 79.86 (23.560)
  Role Functioning Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Role Functioning Score; Cycle 24 Day 1 | 78.89 (16.019) | 83.33 (19.245)
  Role Functioning Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Role Functioning Score; Cycle 25 Day 1 | 77.78 (17.885) | 82.29 (23.936)
  Role Functioning Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Role Functioning Score; Cycle 26 Day 1 | 75 (12.599) | 69.23 (31.066)
  Role Functioning Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Role Functioning Score; Cycle 27 Day 1 | 77.78 (13.608) | 90.48 (16.265)
  Role Functioning Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Role Functioning Score; Cycle 28 Day 1 | 79.17 (15.957) | 97.22 (6.804)
  Role Functioning Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Role Functioning Score; Cycle 29 Day 1 | 75 (9.623) | 96.67 (7.454)
  Role Functioning Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Role Functioning Score; Cycle 30 Day 1 | 87.50 (15.957) | 100
  Role Functioning Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Role Functioning Score; Cycle 31 Day 1 | 66.67 |
  Role Functioning Score; Off-treatment Visit: number analyzed (Participants) | 79 | 74
  Role Functioning Score; Off-treatment Visit | 60.97 (31.790) | 63.51 (31.656)
  Emotional Functioning Score; Baseline | 79.35 (19.704) | 80.06 (19.729)
  Emotional Functioning Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 151
  Emotional Functioning Score; Cycle 2 Day 1 | 79.41 (19.465) | 82.06 (19.167)
  Emotional Functioning Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 141
  Emotional Functioning Score; Cycle 3 Day 1 | 78.47 (21.642) | 82.90 (19.314)
  Emotional Functioning Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 136
  Emotional Functioning Score; Cycle 4 Day 1 | 78.26 (18.854) | 84.19 (18.517)
  Emotional Functioning Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 126
  Emotional Functioning Score; Cycle 5 Day 1 | 75.85 (21.767) | 84.52 (15.766)
  Emotional Functioning Score; Cycle 6 Day 1: number analyzed (Participants) | 121 | 119
  Emotional Functioning Score; Cycle 6 Day 1 | 80.60 (18.703) | 84.38 (18.365)
  Emotional Functioning Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Emotional Functioning Score; Cycle 7 Day 1 | 77.18 (19.571) | 84.29 (16.356)
  Emotional Functioning Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Emotional Functioning Score; Cycle 8 Day 1 | 79.08 (19.744) | 84.88 (18.215)
  Emotional Functioning Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Emotional Functioning Score; Cycle 9 Day 1 | 78.75 (22.127) | 85.96 (17.512)
  Emotional Functioning Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 74
  Emotional Functioning Score; Cycle 10 Day 1 | 80.04 (19.440) | 87.84 (15.433)
  Emotional Functioning Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Emotional Functioning Score; Cycle 11 Day 1 | 82.25 (20.558) | 87.15 (16.247)
  Emotional Functioning Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 60
  Emotional Functioning Score; Cycle 12 Day 1 | 81.51 (19.157) | 86.67 (15.358)
  Emotional Functioning Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Emotional Functioning Score; Cycle 13 Day 1 | 79.32 (17.908) | 87.27 (15.783)
  Emotional Functioning Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Emotional Functioning Score; Cycle 14 Day 1 | 81.35 (16.782) | 87.50 (17.110)
  Emotional Functioning Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Emotional Functioning Score; Cycle 15 Day 1 | 80.30 (18.336) | 87.25 (15.398)
  Emotional Functioning Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Emotional Functioning Score; Cycle 16 Day 1 | 81.50 (17.432) | 87.41 (14.935)
  Emotional Functioning Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Emotional Functioning Score; Cycle 17 Day 1 | 79.63 (19.664) | 87.08 (16.118)
  Emotional Functioning Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Emotional Functioning Score; Cycle 18 Day 1 | 81.90 (15.330) | 86.76 (16.555)
  Emotional Functioning Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Emotional Functioning Score; Cycle 19 Day 1 | 81.17 (15.945) | 84.80 (18.403)
  Emotional Functioning Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Emotional Functioning Score; Cycle 20 Day 1 | 80.25 (17.925) | 86.56 (17.437)
  Emotional Functioning Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Emotional Functioning Score; Cycle 21 Day 1 | 81.73 (15.279) | 88.99 (14.174)
  Emotional Functioning Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Emotional Functioning Score; Cycle 22 Day 1 | 85.09 (16.096) | 89.20 (15.644)
  Emotional Functioning Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Emotional Functioning Score; Cycle 23 Day 1 | 86.67 (15.366) | 87.15 (15.922)
  Emotional Functioning Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Emotional Functioning Score; Cycle 24 Day 1 | 88.89 (14.319) | 87.28 (13.712)
  Emotional Functioning Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Emotional Functioning Score; Cycle 25 Day 1 | 83.33 (18.119) | 90.63 (12.500)
  Emotional Functioning Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Emotional Functioning Score; Cycle 26 Day 1 | 77.08 (23.038) | 85.26 (23.362)
  Emotional Functioning Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Emotional Functioning Score; Cycle 27 Day 1 | 80.56 (16.387) | 95.24 (12.599)
  Emotional Functioning Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Emotional Functioning Score; Cycle 28 Day 1 | 75 (16.667) | 100 (0)
  Emotional Functioning Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Emotional Functioning Score; Cycle 29 Day 1 | 75 (16.667) | 100 (0)
  Emotional Functioning Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Emotional Functioning Score; Cycle 30 Day 1 | 75 (16.667) | 100
  Emotional Functioning Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Emotional Functioning Score; Cycle 31 Day 1 | 66.67 |
  Emotional Functioning Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Emotional Functioning Score; Off-treatment Visit | 69.62 (27.304) | 73.87 (25.145)
  Cognitive Functioning Score; Baseline | 87.91 (15.764) | 89.51 (15.529)
  Cognitive Functioning Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 151
  Cognitive Functioning Score; Cycle 2 Day 1 | 87.15 (15.661) | 88.85 (18.025)
  Cognitive Functioning Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 141
  Cognitive Functioning Score; Cycle 3 Day 1 | 84.45 (19.049) | 87.47 (17.946)
  Cognitive Functioning Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 136
  Cognitive Functioning Score; Cycle 4 Day 1 | 83.58 (19.461) | 90.32 (13.692)
  Cognitive Functioning Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 126
  Cognitive Functioning Score; Cycle 5 Day 1 | 83.99 (17.239) | 87.43 (17.086)
  Cognitive Functioning Score; Cycle 6 Day 1: number analyzed (Participants) | 121 | 119
  Cognitive Functioning Score; Cycle 6 Day 1 | 84.71 (16.886) | 87.68 (18.470)
  Cognitive Functioning Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Cognitive Functioning Score; Cycle 7 Day 1 | 82.40 (18.855) | 87.94 (14.708)
  Cognitive Functioning Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Cognitive Functioning Score; Cycle 8 Day 1 | 81.97 (21.227) | 88.49 (16.380)
  Cognitive Functioning Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Cognitive Functioning Score; Cycle 9 Day 1 | 83.70 (18.084) | 87.68 (17.095)
  Cognitive Functioning Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Cognitive Functioning Score; Cycle 10 Day 1 | 85.39 (17.947) | 90.44 (13.747)
  Cognitive Functioning Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Cognitive Functioning Score; Cycle 11 Day 1 | 84.06 (18.176) | 88.89 (15.824)
  Cognitive Functioning Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 60
  Cognitive Functioning Score; Cycle 12 Day 1 | 85.42 (16.400) | 88.61 (17.758)
  Cognitive Functioning Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Cognitive Functioning Score; Cycle 13 Day 1 | 83.93 (17.685) | 89.70 (12.624)
  Cognitive Functioning Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Cognitive Functioning Score; Cycle 14 Day 1 | 85.71 (18.634) | 87.18 (16.375)
  Cognitive Functioning Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Cognitive Functioning Score; Cycle 15 Day 1 | 84.85 (18.264) | 83.99 (17.308)
  Cognitive Functioning Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Cognitive Functioning Score; Cycle 16 Day 1 | 83.74 (18.062) | 89.36 (13.649)
  Cognitive Functioning Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Cognitive Functioning Score; Cycle 17 Day 1 | 82.87 (18.033) | 89.58 (14.465)
  Cognitive Functioning Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Cognitive Functioning Score; Cycle 18 Day 1 | 83.87 (17.994) | 90.20 (15.417)
  Cognitive Functioning Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Cognitive Functioning Score; Cycle 19 Day 1 | 80.25 (18.511) | 89.22 (14.727)
  Cognitive Functioning Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Cognitive Functioning Score; Cycle 20 Day 1 | 82.10 (17.250) | 91.94 (12.073)
  Cognitive Functioning Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Cognitive Functioning Score; Cycle 21 Day 1 | 81.41 (19.623) | 88.10 (12.715)
  Cognitive Functioning Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Cognitive Functioning Score; Cycle 22 Day 1 | 88.60 (14.754) | 90.12 (12.454)
  Cognitive Functioning Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Cognitive Functioning Score; Cycle 23 Day 1 | 83.33 (16.667) | 88.19 (14.311)
  Cognitive Functioning Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Cognitive Functioning Score; Cycle 24 Day 1 | 84.44 (16.019) | 92.11 (8.550)
  Cognitive Functioning Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Cognitive Functioning Score; Cycle 25 Day 1 | 84.72 (15.006) | 98.96 (4.167)
  Cognitive Functioning Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Cognitive Functioning Score; Cycle 26 Day 1 | 89.58 (12.400) | 92.31 (11.004)
  Cognitive Functioning Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Cognitive Functioning Score; Cycle 27 Day 1 | 83.33 (14.907) | 95.24 (12.599)
  Cognitive Functioning Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Cognitive Functioning Score; Cycle 28 Day 1 | 91.67 (9.623) | 100 (0)
  Cognitive Functioning Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Cognitive Functioning Score; Cycle 29 Day 1 | 91.67 (9.623) | 100 (0)
  Cognitive Functioning Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Cognitive Functioning Score; Cycle 30 Day 1 | 87.50 (15.957) | 100
  Cognitive Functioning Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Cognitive Functioning Score; Cycle 31 Day 1 | 83.33 |
  Cognitive Functioning Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Cognitive Functioning Score; Off-treatment Visit | 75.21 (25.846) | 80.41 (23.304)
  Social Functioning Score; Baseline | 77.29 (25.678) | 78.29 (27.243)
  Social Functioning Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 151
  Social Functioning Score; Cycle 2 Day 1 | 73.46 (25.386) | 77.15 (27.190)
  Social Functioning Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 141
  Social Functioning Score; Cycle 3 Day 1 | 72.04 (26.229) | 77.19 (25.309)
  Social Functioning Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 136
  Social Functioning Score; Cycle 4 Day 1 | 71.43 (24.837) | 77.33 (25.311)
  Social Functioning Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 126
  Social Functioning Score; Cycle 5 Day 1 | 71.78 (25.589) | 79.63 (23.934)
  Social Functioning Score; Cycle 6 Day 1: number analyzed (Participants) | 121 | 119
  Social Functioning Score; Cycle 6 Day 1 | 70.80 (26.812) | 78.71 (25.758)
  Social Functioning Score; Cycle 7 Day 1: number analyzed (Participants) | 106 | 105
  Social Functioning Score; Cycle 7 Day 1 | 71.70 (26.544) | 77.30 (24.691)
  Social Functioning Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Social Functioning Score; Cycle 8 Day 1 | 70.24 (28.139) | 79.04 (24.565)
  Social Functioning Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Social Functioning Score; Cycle 9 Day 1 | 72.16 (25.946) | 78.62 (20.573)
  Social Functioning Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 74
  Social Functioning Score; Cycle 10 Day 1 | 72.43 (28.156) | 85.14 (19.422)
  Social Functioning Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Social Functioning Score; Cycle 11 Day 1 | 73.91 (25.801) | 85.19 (19.086)
  Social Functioning Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 60
  Social Functioning Score; Cycle 12 Day 1 | 76.56 (24.073) | 83.89 (23.161)
  Social Functioning Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Social Functioning Score; Cycle 13 Day 1 | 72.92 (23.476) | 83.94 (21.508)
  Social Functioning Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Social Functioning Score; Cycle 14 Day 1 | 72.79 (22.997) | 83.97 (19.792)
  Social Functioning Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Social Functioning Score; Cycle 15 Day 1 | 72.73 (25.942) | 81.37 (22.273)
  Social Functioning Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 46
  Social Functioning Score; Cycle 16 Day 1 | 73.17 (24.403) | 80.80 (22.489)
  Social Functioning Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Social Functioning Score; Cycle 17 Day 1 | 70.37 (22.222) | 80.42 (24.134)
  Social Functioning Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Social Functioning Score; Cycle 18 Day 1 | 76.88 (20.493) | 82.84 (21.116)
  Social Functioning Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Social Functioning Score; Cycle 19 Day 1 | 74.07 (22.329) | 80.88 (25.667)
  Social Functioning Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Social Functioning Score; Cycle 20 Day 1 | 75.31 (24.183) | 81.72 (22.092)
  Social Functioning Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Social Functioning Score; Cycle 21 Day 1 | 73.72 (18.362) | 82.14 (24.398)
  Social Functioning Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Social Functioning Score; Cycle 22 Day 1 | 79.82 (17.194) | 82.10 (20.634)
  Social Functioning Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Social Functioning Score; Cycle 23 Day 1 | 82.22 (18.330) | 83.33 (22.522)
  Social Functioning Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Social Functioning Score; Cycle 24 Day 1 | 83.33 (17.817) | 84.21 (19.621)
  Social Functioning Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Social Functioning Score; Cycle 25 Day 1 | 87.50 (12.563) | 84.38 (18.727)
  Social Functioning Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Social Functioning Score; Cycle 26 Day 1 | 83.33 (15.430) | 76.92 (31.578)
  Social Functioning Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Social Functioning Score; Cycle 27 Day 1 | 80.56 (12.546) | 95.24 (12.599)
  Social Functioning Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Social Functioning Score; Cycle 28 Day 1 | 83.33 (19.245) | 100 (0)
  Social Functioning Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Social Functioning Score; Cycle 29 Day 1 | 79.17 (15.957) | 100 (0)
  Social Functioning Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Social Functioning Score; Cycle 30 Day 1 | 70.83 (8.333) | 100
  Social Functioning Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Social Functioning Score; Cycle 31 Day 1 | 100 |
  Social Functioning Score; Off-treatment Visit: number analyzed (Participants) | 80 | 73
  Social Functioning Score; Off-treatment Visit | 64.58 (31.419) | 66.89 (32.453)
  Fatigue Score; Baseline | 31.32 (21.379) | 31.76 (25.224)
  Fatigue Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 150
  Fatigue Score; Cycle 2 Day 1 | 39.21 (22.171) | 36.74 (23.665)
  Fatigue Score; Cycle 3 Day 1: number analyzed (Participants) | 148 | 142
  Fatigue Score; Cycle 3 Day 1 | 40.09 (24.095) | 36.62 (24.031)
  Fatigue Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 137
  Fatigue Score; Cycle 4 Day 1 | 40.21 (23.504) | 32.68 (23.829)
  Fatigue Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 127
  Fatigue Score; Cycle 5 Day 1 | 37.54 (23.329) | 35.17 (22.431)
  Fatigue Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Fatigue Score; Cycle 6 Day 1 | 38.80 (23.246) | 33.19 (23.696)
  Fatigue Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Fatigue Score; Cycle 7 Day 1 | 38.06 (21.850) | 30.79 (21.859)
  Fatigue Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Fatigue Score; Cycle 8 Day 1 | 36.14 (22.852) | 30.81 (23.268)
  Fatigue Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Fatigue Score; Cycle 9 Day 1 | 35.90 (21.281) | 30.80 (21.293)
  Fatigue Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Fatigue Score; Cycle 10 Day 1 | 34.57 (22.635) | 27.11 (20.278)
  Fatigue Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Fatigue Score; Cycle 11 Day 1 | 32.37 (20.851) | 27.46 (22.788)
  Fatigue Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Fatigue Score; Cycle 12 Day 1 | 32.82 (20.264) | 23.48 (21.302)
  Fatigue Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Fatigue Score; Cycle 13 Day 1 | 35.52 (18.882) | 25.05 (21.300)
  Fatigue Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Fatigue Score; Cycle 14 Day 1 | 30.84 (21.429) | 25.58 (20.276)
  Fatigue Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Fatigue Score; Cycle 15 Day 1 | 28.03 (20.682) | 28.98 (23.315)
  Fatigue Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Fatigue Score; Cycle 16 Day 1 | 33.33 (22.361) | 25.53 (20.581)
  Fatigue Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Fatigue Score; Cycle 17 Day 1 | 33.33 (21.902) | 25 (20.090)
  Fatigue Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Fatigue Score; Cycle 18 Day 1 | 34.05 (22.024) | 24.84 (19.546)
  Fatigue Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Fatigue Score; Cycle 19 Day 1 | 37.04 (23.061) | 27.45 (22.595)
  Fatigue Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Fatigue Score; Cycle 20 Day 1 | 34.57 (19.812) | 27.24 (22.192)
  Fatigue Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Fatigue Score; Cycle 21 Day 1 | 34.19 (20.828) | 23.02 (17.088)
  Fatigue Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Fatigue Score; Cycle 22 Day 1 | 26.32 (18.596) | 26.75 (20.033)
  Fatigue Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Fatigue Score; Cycle 23 Day 1 | 26.67 (20.053) | 29.17 (21.934)
  Fatigue Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Fatigue Score; Cycle 24 Day 1 | 28.15 (20.082) | 26.90 (17.496)
  Fatigue Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Fatigue Score; Cycle 25 Day 1 | 33.33 (19.534) | 25.69 (19.338)
  Fatigue Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Fatigue Score; Cycle 26 Day 1 | 26.39 (17.755) | 37.61 (28.160)
  Fatigue Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Fatigue Score; Cycle 27 Day 1 | 27.78 (16.851) | 20.63 (20.716)
  Fatigue Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Fatigue Score; Cycle 28 Day 1 | 22.22 (15.713) | 16.67 (19.563)
  Fatigue Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Fatigue Score; Cycle 29 Day 1 | 22.22 (15.713) | 15.56 (14.907)
  Fatigue Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Fatigue Score; Cycle 30 Day 1 | 25 (16.667) | 11.11
  Fatigue Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Fatigue Score; Cycle 31 Day 1 | 33.33 |
  Fatigue Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Fatigue Score; Off-treatment Visit | 43.47 (28.173) | 38.89 (28.977)
  Nausea and Vomiting Score; Baseline | 7.60 (17.265) | 6.28 (14.510)
  Nausea and Vomiting Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 150
  Nausea and Vomiting Score; Cycle 2 Day 1 | 11.50 (18.229) | 9.56 (17.943)
  Nausea and Vomiting Score; Cycle 3 Day 1: number analyzed (Participants) | 148 | 142
  Nausea and Vomiting Score; Cycle 3 Day 1 | 14.86 (24.057) | 9.74 (18.219)
  Nausea and Vomiting Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 137
  Nausea and Vomiting Score; Cycle 4 Day 1 | 15.80 (21.386) | 12.17 (18.906)
  Nausea and Vomiting Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 127
  Nausea and Vomiting Score; Cycle 5 Day 1 | 12.07 (17.017) | 11.42 (18.270)
  Nausea and Vomiting Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Nausea and Vomiting Score; Cycle 6 Day 1 | 12.74 (19.215) | 10.14 (18.996)
  Nausea and Vomiting Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Nausea and Vomiting Score; Cycle 7 Day 1 | 12.46 (18.612) | 8.57 (13.696)
  Nausea and Vomiting Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Nausea and Vomiting Score; Cycle 8 Day 1 | 13.10 (21.836) | 10.14 (15.508)
  Nausea and Vomiting Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Nausea and Vomiting Score; Cycle 9 Day 1 | 12.27 (20.005) | 9.96 (17.306)
  Nausea and Vomiting Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Nausea and Vomiting Score; Cycle 10 Day 1 | 15.02 (22.299) | 7.78 (16.287)
  Nausea and Vomiting Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Nausea and Vomiting Score; Cycle 11 Day 1 | 11.11 (18.002) | 8.69 (15.394)
  Nausea and Vomiting Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Nausea and Vomiting Score; Cycle 12 Day 1 | 12.82 (19.042) | 6.99 (14.645)
  Nausea and Vomiting Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Nausea and Vomiting Score; Cycle 13 Day 1 | 12.20 (18.934) | 6.97 (13.867)
  Nausea and Vomiting Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Nausea and Vomiting Score; Cycle 14 Day 1 | 14.97 (21.849) | 7.55 (16.527)
  Nausea and Vomiting Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Nausea and Vomiting Score; Cycle 15 Day 1 | 14.02 (20.631) | 8.82 (15.038)
  Nausea and Vomiting Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Nausea and Vomiting Score; Cycle 16 Day 1 | 11.38 (19.874) | 9.22 (15.467)
  Nausea and Vomiting Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Nausea and Vomiting Score; Cycle 17 Day 1 | 14.35 (22.940) | 5 (13.183)
  Nausea and Vomiting Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Nausea and Vomiting Score; Cycle 18 Day 1 | 10.75 (22.587) | 9.31 (15.457)
  Nausea and Vomiting Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Nausea and Vomiting Score; Cycle 19 Day 1 | 16.67 (27.347) | 7.35 (15.457)
  Nausea and Vomiting Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Nausea and Vomiting Score; Cycle 20 Day 1 | 16.67 (23.113) | 10.22 (15.915)
  Nausea and Vomiting Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Nausea and Vomiting Score; Cycle 21 Day 1 | 12.82 (20.714) | 7.74 (12.408)
  Nausea and Vomiting Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Nausea and Vomiting Score; Cycle 22 Day 1 | 7.02 (11.541) | 8.64 (13.374)
  Nausea and Vomiting Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Nausea and Vomiting Score; Cycle 23 Day 1 | 5.56 (12.062) | 6.25 (11.849)
  Nausea and Vomiting Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Nausea and Vomiting Score; Cycle 24 Day 1 | 6.67 (13.801) | 7.89 (17.004)
  Nausea and Vomiting Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Nausea and Vomiting Score; Cycle 25 Day 1 | 13.89 (21.122) | 2.08 (8.333)
  Nausea and Vomiting Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Nausea and Vomiting Score; Cycle 26 Day 1 | 4.17 (7.715) | 14.10 (24.387)
  Nausea and Vomiting Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Nausea and Vomiting Score; Cycle 27 Day 1 | 5.56 (13.608) | 16.67 (28.868)
  Nausea and Vomiting Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Nausea and Vomiting Score; Cycle 28 Day 1 | 12.50 (15.957) | 8.33 (20.412)
  Nausea and Vomiting Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Nausea and Vomiting Score; Cycle 29 Day 1 | 16.67 (13.608) | 0 (0)
  Nausea and Vomiting Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Nausea and Vomiting Score; Cycle 30 Day 1 | 8.33 (16.667) | 0
  Nausea and Vomiting Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Nausea and Vomiting Score; Cycle 31 Day 1 | 16.67 |
  Nausea and Vomiting Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Nausea and Vomiting Score; Off-treatment Visit | 13.33 (22.564) | 6.76 (13.207)
  Pain Score; Baseline | 23.39 (25.410) | 23.77 (26.323)
  Pain Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 151
  Pain Score; Cycle 2 Day 1 | 26.79 (25.850) | 27.04 (23.862)
  Pain Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 142
  Pain Score; Cycle 3 Day 1 | 27.63 (24.103) | 25 (24.046)
  Pain Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 137
  Pain Score; Cycle 4 Day 1 | 26.67 (24.788) | 22.87 (21.486)
  Pain Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 127
  Pain Score; Cycle 5 Day 1 | 29.04 (26.805) | 22.97 (22.314)
  Pain Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Pain Score; Cycle 6 Day 1 | 26.29 (24.887) | 22.50 (25.716)
  Pain Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Pain Score; Cycle 7 Day 1 | 28.04 (23.189) | 23.65 (22.142)
  Pain Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 97
  Pain Score; Cycle 8 Day 1 | 27.38 (23.722) | 23.20 (24.949)
  Pain Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Pain Score; Cycle 9 Day 1 | 27.11 (23.393) | 21.01 (20.053)
  Pain Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Pain Score; Cycle 10 Day 1 | 26.95 (22.603) | 19.33 (18.792)
  Pain Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Pain Score; Cycle 11 Day 1 | 27.29 (22.319) | 18.06 (20.508)
  Pain Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Pain Score; Cycle 12 Day 1 | 26.41 (21.018) | 18.55 (19.814)
  Pain Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Pain Score; Cycle 13 Day 1 | 24.40 (20.092) | 18.48 (20.203)
  Pain Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Pain Score; Cycle 14 Day 1 | 22.11 (22.666) | 16.04 (19.601)
  Pain Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 53
  Pain Score; Cycle 15 Day 1 | 24.24 (23.966) | 17.65 (18.078)
  Pain Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Pain Score; Cycle 16 Day 1 | 29.67 (25.417) | 18.44 (20.628)
  Pain Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Pain Score; Cycle 17 Day 1 | 27.78 (25.198) | 17.50 (19.954)
  Pain Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Pain Score; Cycle 18 Day 1 | 25.27 (20.125) | 16.67 (18.803)
  Pain Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Pain Score; Cycle 19 Day 1 | 31.48 (23.266) | 19.61 (22.274)
  Pain Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Pain Score; Cycle 20 Day 1 | 29.63 (23.266) | 19.35 (21.558)
  Pain Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Pain Score; Cycle 21 Day 1 | 26.92 (23.131) | 17.86 (21.721)
  Pain Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Pain Score; Cycle 22 Day 1 | 23.68 (17.843) | 22.84 (24.085)
  Pain Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Pain Score; Cycle 23 Day 1 | 21.11 (14.729) | 18.06 (23.527)
  Pain Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Pain Score; Cycle 24 Day 1 | 22.22 (20.574) | 14.91 (19.160)
  Pain Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Pain Score; Cycle 25 Day 1 | 27.78 (23.925) | 15.63 (19.691)
  Pain Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Pain Score; Cycle 26 Day 1 | 27.08 (21.708) | 21.79 (27.542)
  Pain Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Pain Score; Cycle 27 Day 1 | 25 (20.412) | 11.90 (24.934)
  Pain Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Pain Score; Cycle 28 Day 1 | 25 (21.517) | 2.78 (6.804)
  Pain Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Pain Score; Cycle 29 Day 1 | 25 (21.517) | 6.67 (14.907)
  Pain Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Pain Score; Cycle 30 Day 1 | 25 (16.667) | 0
  Pain Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Pain Score; Cycle 31 Day 1 | 33.33 |
  Pain Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Pain Score; Off-treatment Visit | 28.33 (27.354) | 27.70 (28.171)
  Dyspnea Score; Baseline: number analyzed (Participants) | 170 | 162
  Dyspnea Score; Baseline | 21.18 (25.562) | 22.22 (26.006)
  Dyspnea Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 150
  Dyspnea Score; Cycle 2 Day 1 | 18.90 (24.248) | 19.56 (23.865)
  Dyspnea Score; Cycle 3 Day 1: number analyzed (Participants) | 147 | 142
  Dyspnea Score; Cycle 3 Day 1 | 20.63 (24.155) | 19.72 (23.871)
  Dyspnea Score; Cycle 4 Day 1: number analyzed (Participants) | 134 | 137
  Dyspnea Score; Cycle 4 Day 1 | 19.90 (24.224) | 17.52 (20.643)
  Dyspnea Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 127
  Dyspnea Score; Cycle 5 Day 1 | 19.16 (23.201) | 15.75 (20.925)
  Dyspnea Score; Cycle 6 Day 1: number analyzed (Participants) | 122 | 120
  Dyspnea Score; Cycle 6 Day 1 | 16.67 (21.104) | 18.89 (23.957)
  Dyspnea Score; Cycle 7 Day 1: number analyzed (Participants) | 105 | 105
  Dyspnea Score; Cycle 7 Day 1 | 19.37 (23.922) | 15.87 (21.728)
  Dyspnea Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Dyspnea Score; Cycle 8 Day 1 | 19.24 (23.489) | 14.09 (20.319)
  Dyspnea Score; Cycle 9 Day 1: number analyzed (Participants) | 90 | 92
  Dyspnea Score; Cycle 9 Day 1 | 15.93 (20.740) | 14.49 (21.712)
  Dyspnea Score; Cycle 10 Day 1: number analyzed (Participants) | 80 | 75
  Dyspnea Score; Cycle 10 Day 1 | 17.92 (21.832) | 11.56 (19.369)
  Dyspnea Score; Cycle 11 Day 1: number analyzed (Participants) | 68 | 71
  Dyspnea Score; Cycle 11 Day 1 | 18.63 (23.310) | 15.02 (23.764)
  Dyspnea Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 62
  Dyspnea Score; Cycle 12 Day 1 | 13.54 (21.998) | 12.90 (22.057)
  Dyspnea Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Dyspnea Score; Cycle 13 Day 1 | 13.69 (20.867) | 10.91 (20.341)
  Dyspnea Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Dyspnea Score; Cycle 14 Day 1 | 15.65 (21.626) | 10.69 (20.437)
  Dyspnea Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Dyspnea Score; Cycle 15 Day 1 | 15.15 (19.628) | 12.42 (21.040)
  Dyspnea Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Dyspnea Score; Cycle 16 Day 1 | 16.26 (22.512) | 9.93 (16.904)
  Dyspnea Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Dyspnea Score; Cycle 17 Day 1 | 15.74 (20.293) | 10 (20.255)
  Dyspnea Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Dyspnea Score; Cycle 18 Day 1 | 16.13 (20.854) | 10.78 (17.829)
  Dyspnea Score; Cycle 19 Day 1: number analyzed (Participants) | 26 | 34
  Dyspnea Score; Cycle 19 Day 1 | 15.38 (21.563) | 9.80 (17.465)
  Dyspnea Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Dyspnea Score; Cycle 20 Day 1 | 23.46 (20.286) | 11.83 (16.212)
  Dyspnea Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Dyspnea Score; Cycle 21 Day 1 | 15.38 (16.946) | 7.14 (13.929)
  Dyspnea Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Dyspnea Score; Cycle 22 Day 1 | 17.54 (20.393) | 12.35 (18.829)
  Dyspnea Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Dyspnea Score; Cycle 23 Day 1 | 13.33 (21.082) | 11.11 (18.822)
  Dyspnea Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Dyspnea Score; Cycle 24 Day 1 | 20 (21.082) | 12.28 (16.520)
  Dyspnea Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Dyspnea Score; Cycle 25 Day 1 | 22.22 (29.588) | 8.33 (14.907)
  Dyspnea Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Dyspnea Score; Cycle 26 Day 1 | 16.67 (17.817) | 15.38 (22.008)
  Dyspnea Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Dyspnea Score; Cycle 27 Day 1 | 11.11 (17.213) | 14.29 (17.817)
  Dyspnea Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Dyspnea Score; Cycle 28 Day 1 | 16.67 (19.245) | 16.67 (18.257)
  Dyspnea Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Dyspnea Score; Cycle 29 Day 1 | 25 (16.667) | 20 (18.257)
  Dyspnea Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Dyspnea Score; Cycle 30 Day 1 | 16.67 (19.245) | 0
  Dyspnea Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Dyspnea Score; Cycle 31 Day 1 | 33.33 |
  Dyspnea Score; Off-treatment Visit: number analyzed (Participants) | 77 | 74
  Dyspnea Score; Off-treatment Visit | 24.68 (27.254) | 21.62 (28.898)
  Insomnia Score; Baseline: number analyzed (Participants) | 169 | 162
  Insomnia Score; Baseline | 23.08 (26.972) | 22.84 (27.671)
  Insomnia Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 149
  Insomnia Score; Cycle 2 Day 1 | 26.11 (27.038) | 19.91 (25.386)
  Insomnia Score; Cycle 3 Day 1: number analyzed (Participants) | 147 | 142
  Insomnia Score; Cycle 3 Day 1 | 30.39 (29.435) | 23 (25.477)
  Insomnia Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 137
  Insomnia Score; Cycle 4 Day 1 | 26.57 (28.057) | 20.19 (24.036)
  Insomnia Score; Cycle 5 Day 1: number analyzed (Participants) | 126 | 127
  Insomnia Score; Cycle 5 Day 1 | 23.02 (26.487) | 22.05 (24.205)
  Insomnia Score; Cycle 6 Day 1: number analyzed (Participants) | 122 | 120
  Insomnia Score; Cycle 6 Day 1 | 24.86 (26.955) | 17.50 (22.019)
  Insomnia Score; Cycle 7 Day 1: number analyzed (Participants) | 105 | 105
  Insomnia Score; Cycle 7 Day 1 | 25.08 (27.651) | 20 (25.149)
  Insomnia Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Insomnia Score; Cycle 8 Day 1 | 26.46 (28.843) | 19.59 (25.346)
  Insomnia Score; Cycle 9 Day 1: number analyzed (Participants) | 90 | 92
  Insomnia Score; Cycle 9 Day 1 | 25.56 (27.392) | 16.67 (21.255)
  Insomnia Score; Cycle 10 Day 1: number analyzed (Participants) | 80 | 75
  Insomnia Score; Cycle 10 Day 1 | 24.58 (25.844) | 18.22 (22.789)
  Insomnia Score; Cycle 11 Day 1: number analyzed (Participants) | 68 | 71
  Insomnia Score; Cycle 11 Day 1 | 24.02 (26.918) | 17.37 (24.468)
  Insomnia Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 62
  Insomnia Score; Cycle 12 Day 1 | 23.44 (23.518) | 13.98 (22.216)
  Insomnia Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Insomnia Score; Cycle 13 Day 1 | 21.43 (21.489) | 13.33 (21.849)
  Insomnia Score; Cycle 14 Day 1: number analyzed (Participants) | 48 | 53
  Insomnia Score; Cycle 14 Day 1 | 18.06 (23.778) | 11.95 (21.774)
  Insomnia Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 50
  Insomnia Score; Cycle 15 Day 1 | 18.94 (20.832) | 16 (23.561)
  Insomnia Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Insomnia Score; Cycle 16 Day 1 | 20.33 (20.921) | 14.89 (21.768)
  Insomnia Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Insomnia Score; Cycle 17 Day 1 | 17.59 (16.877) | 13.33 (21.082)
  Insomnia Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Insomnia Score; Cycle 18 Day 1 | 27.96 (25.958) | 11.76 (19.903)
  Insomnia Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Insomnia Score; Cycle 19 Day 1 | 24.69 (25.474) | 13.73 (21.893)
  Insomnia Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Insomnia Score; Cycle 20 Day 1 | 25.93 (25.036) | 12.90 (20.507)
  Insomnia Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Insomnia Score; Cycle 21 Day 1 | 23.08 (27.919) | 10.71 (18.265)
  Insomnia Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Insomnia Score; Cycle 22 Day 1 | 21.05 (19.909) | 6.17 (16.111)
  Insomnia Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Insomnia Score; Cycle 23 Day 1 | 26.67 (22.537) | 11.11 (23.399)
  Insomnia Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Insomnia Score; Cycle 24 Day 1 | 24.44 (26.627) | 12.28 (19.909)
  Insomnia Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Insomnia Score; Cycle 25 Day 1 | 16.67 (17.408) | 12.50 (20.638)
  Insomnia Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Insomnia Score; Cycle 26 Day 1 | 16.67 (17.817) | 20.51 (32.026)
  Insomnia Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Insomnia Score; Cycle 27 Day 1 | 22.22 (17.213) | 9.52 (16.265)
  Insomnia Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Insomnia Score; Cycle 28 Day 1 | 25 (16.667) | 11.11 (17.213)
  Insomnia Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Insomnia Score; Cycle 29 Day 1 | 25 (16.667) | 13.33 (18.257)
  Insomnia Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Insomnia Score; Cycle 30 Day 1 | 25 (16.667) | 0
  Insomnia Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Insomnia Score; Cycle 31 Day 1 | 33.33 |
  Insomnia Score; Off-treatment Visit: number analyzed (Participants) | 78 | 74
  Insomnia Score; Off-treatment Visit | 32.05 (32.430) | 28.83 (31.850)
  Appetite Loss Score; Baseline | 15.79 (24.606) | 18.31 (27.060)
  Appetite Loss Score; Cycle 2 Day 1: number analyzed (Participants) | 158 | 150
  Appetite Loss Score; Cycle 2 Day 1 | 26.79 (31.129) | 27.56 (32.020)
  Appetite Loss Score; Cycle 3 Day 1: number analyzed (Participants) | 147 | 142
  Appetite Loss Score; Cycle 3 Day 1 | 31.97 (31.905) | 29.81 (31.687)
  Appetite Loss Score; Cycle 4 Day 1: number analyzed (Participants) | 134 | 137
  Appetite Loss Score; Cycle 4 Day 1 | 32.09 (31.239) | 30.90 (32.749)
  Appetite Loss Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 125
  Appetite Loss Score; Cycle 5 Day 1 | 30.47 (29.881) | 30.67 (32.129)
  Appetite Loss Score; Cycle 6 Day 1: number analyzed (Participants) | 123 | 120
  Appetite Loss Score; Cycle 6 Day 1 | 30.35 (31.365) | 26.11 (29.996)
  Appetite Loss Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Appetite Loss Score; Cycle 7 Day 1 | 29.28 (31.956) | 26.98 (28.154)
  Appetite Loss Score; Cycle 8 Day 1: number analyzed (Participants) | 98 | 96
  Appetite Loss Score; Cycle 8 Day 1 | 29.25 (31.483) | 25.00 (26.491)
  Appetite Loss Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Appetite Loss Score; Cycle 9 Day 1 | 29.30 (30.565) | 25.36 (27.678)
  Appetite Loss Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Appetite Loss Score; Cycle 10 Day 1 | 27.57 (29.716) | 22.22 (22.815)
  Appetite Loss Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Appetite Loss Score; Cycle 11 Day 1 | 24.15 (27.938) | 22.07 (26.988)
  Appetite Loss Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Appetite Loss Score; Cycle 12 Day 1 | 22.05 (24.493) | 18.82 (25.336)
  Appetite Loss Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 54
  Appetite Loss Score; Cycle 13 Day 1 | 23.21 (25.362) | 17.28 (21.221)
  Appetite Loss Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  Appetite Loss Score; Cycle 14 Day 1 | 19.73 (24.456) | 17.61 (24.111)
  Appetite Loss Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Appetite Loss Score; Cycle 15 Day 1 | 17.42 (23.282) | 24.18 (30.608)
  Appetite Loss Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Appetite Loss Score; Cycle 16 Day 1 | 23.58 (27.125) | 22.70 (27.014)
  Appetite Loss Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Appetite Loss Score; Cycle 17 Day 1 | 20.37 (21.496) | 22.50 (25.473)
  Appetite Loss Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 33
  Appetite Loss Score; Cycle 18 Day 1 | 19.35 (22.401) | 22.22 (24.533)
  Appetite Loss Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Appetite Loss Score; Cycle 19 Day 1 | 19.75 (23.130) | 20.59 (25.969)
  Appetite Loss Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Appetite Loss Score; Cycle 20 Day 1 | 23.46 (25.844) | 21.51 (30.488)
  Appetite Loss Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Appetite Loss Score; Cycle 21 Day 1 | 23.08 (20.590) | 15.48 (21.242)
  Appetite Loss Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Appetite Loss Score; Cycle 22 Day 1 | 17.54 (20.393) | 17.28 (25.099)
  Appetite Loss Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Appetite Loss Score; Cycle 23 Day 1 | 17.78 (24.774) | 20.83 (27.474)
  Appetite Loss Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Appetite Loss Score; Cycle 24 Day 1 | 13.33 (24.560) | 15.79 (25.744)
  Appetite Loss Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Appetite Loss Score; Cycle 25 Day 1 | 19.44 (22.285) | 18.75 (29.736)
  Appetite Loss Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Appetite Loss Score; Cycle 26 Day 1 | 29.17 (27.817) | 23.08 (34.385)
  Appetite Loss Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Appetite Loss Score; Cycle 27 Day 1 | 16.67 (18.257) | 9.52 (16.265)
  Appetite Loss Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Appetite Loss Score; Cycle 28 Day 1 | 8.33 (16.667) | 11.11 (17.213)
  Appetite Loss Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Appetite Loss Score; Cycle 29 Day 1 | 16.67 (19.245) | 0 (0)
  Appetite Loss Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Appetite Loss Score; Cycle 30 Day 1 | 8.33 (16.667) | 0
  Appetite Loss Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Appetite Loss Score; Cycle 31 Day 1 | 0 |
  Appetite Loss Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Appetite Loss Score; Off-treatment Visit | 29.58 (31.820) | 25.23 (32.082)
  Constipation Score; Baseline | 15.98 (24.876) | 12.55 (23.501)
  Constipation Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 150
  Constipation Score; Cycle 2 Day 1 | 10.40 (20.274) | 11.11 (21.035)
  Constipation Score; Cycle 3 Day 1: number analyzed (Participants) | 147 | 142
  Constipation Score; Cycle 3 Day 1 | 9.52 (20.644) | 10.80 (20.456)
  Constipation Score; Cycle 4 Day 1: number analyzed (Participants) | 135 | 136
  Constipation Score; Cycle 4 Day 1 | 11.11 (21.930) | 9.80 (19.081)
  Constipation Score; Cycle 5 Day 1: number analyzed (Participants) | 128 | 125
  Constipation Score; Cycle 5 Day 1 | 12.24 (20.438) | 9.87 (19.411)
  Constipation Score; Cycle 6 Day 1: number analyzed (Participants) | 122 | 118
  Constipation Score; Cycle 6 Day 1 | 8.47 (16.905) | 8.47 (19.090)
  Constipation Score; Cycle 7 Day 1: number analyzed (Participants) | 106 | 103
  Constipation Score; Cycle 7 Day 1 | 11.01 (22.874) | 7.44 (16.785)
  Constipation Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Constipation Score; Cycle 8 Day 1 | 9.62 (18.608) | 7.22 (14.614)
  Constipation Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Constipation Score; Cycle 9 Day 1 | 6.23 (15.644) | 9.42 (19.967)
  Constipation Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Constipation Score; Cycle 10 Day 1 | 6.58 (13.354) | 8.00 (18.042)
  Constipation Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  Constipation Score; Cycle 11 Day 1 | 6.76 (15.739) | 7.98 (18.227)
  Constipation Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 62
  Constipation Score; Cycle 12 Day 1 | 5.64 (13.906) | 9.68 (18.492)
  Constipation Score; Cycle 13 Day 1: number analyzed (Participants) | 55 | 55
  Constipation Score; Cycle 13 Day 1 | 3.64 (12.294) | 9.09 (18.653)
  Constipation Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Constipation Score; Cycle 14 Day 1 | 5.44 (14.186) | 7.69 (16.978)
  Constipation Score; Cycle 15 Day 1: number analyzed (Participants) | 43 | 50
  Constipation Score; Cycle 15 Day 1 | 5.43 (17.714) | 9.33 (19.095)
  Constipation Score; Cycle 16 Day 1: number analyzed (Participants) | 39 | 47
  Constipation Score; Cycle 16 Day 1 | 5.98 (16.879) | 9.93 (18.277)
  Constipation Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Constipation Score; Cycle 17 Day 1 | 11.11 (22.537) | 5.00 (12.054)
  Constipation Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Constipation Score; Cycle 18 Day 1 | 7.53 (14.167) | 7.84 (16.532)
  Constipation Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Constipation Score; Cycle 19 Day 1 | 9.88 (18.057) | 9.80 (20.969)
  Constipation Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Constipation Score; Cycle 20 Day 1 | 8.64 (17.523) | 8.60 (22.718)
  Constipation Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Constipation Score; Cycle 21 Day 1 | 8.97 (17.783) | 7.14 (16.623)
  Constipation Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Constipation Score; Cycle 22 Day 1 | 7.02 (13.962) | 7.41 (19.245)
  Constipation Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Constipation Score; Cycle 23 Day 1 | 6.67 (13.801) | 11.11 (21.234)
  Constipation Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Constipation Score; Cycle 24 Day 1 | 4.44 (17.213) | 8.77 (21.779)
  Constipation Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Constipation Score; Cycle 25 Day 1 | 5.56 (12.975) | 18.75 (29.736)
  Constipation Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Constipation Score; Cycle 26 Day 1 | 8.33 (15.430) | 15.38 (25.875)
  Constipation Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Constipation Score; Cycle 27 Day 1 | 16.67 (27.889) | 0 (0)
  Constipation Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Constipation Score; Cycle 28 Day 1 | 25.00 (31.914) | 0 (0)
  Constipation Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Constipation Score; Cycle 29 Day 1 | 25.00 (31.914) | 0 (0)
  Constipation Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Constipation Score; Cycle 30 Day 1 | 16.67 (33.333) | 0
  Constipation Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Constipation Score; Cycle 31 Day 1 | 33.33 |
  Constipation Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Constipation Score; Off-treatment Visit | 13.33 (23.481) | 12.61 (21.863)
  Diarrhea Score; Baseline | 6.43 (15.045) | 6.79 (15.823)
  Diarrhea Score; Cycle 2 Day 1: number analyzed (Participants) | 157 | 151
  Diarrhea Score; Cycle 2 Day 1 | 22.29 (29.572) | 17.66 (26.333)
  Diarrhea Score; Cycle 3 Day 1: number analyzed (Participants) | 149 | 141
  Diarrhea Score; Cycle 3 Day 1 | 32.21 (30.858) | 27.19 (32.023)
  Diarrhea Score; Cycle 4 Day 1: number analyzed (Participants) | 133 | 136
  Diarrhea Score; Cycle 4 Day 1 | 35.59 (33.634) | 29.41 (28.991)
  Diarrhea Score; Cycle 5 Day 1: number analyzed (Participants) | 127 | 125
  Diarrhea Score; Cycle 5 Day 1 | 28.61 (28.085) | 29.33 (29.207)
  Diarrhea Score; Cycle 6 Day 1: number analyzed (Participants) | 121 | 119
  Diarrhea Score; Cycle 6 Day 1 | 31.96 (30.550) | 26.89 (27.541)
  Diarrhea Score; Cycle 7 Day 1: number analyzed (Participants) | 107 | 105
  Diarrhea Score; Cycle 7 Day 1 | 33.64 (31.885) | 31.75 (27.881)
  Diarrhea Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Diarrhea Score; Cycle 8 Day 1 | 29.55 (28.818) | 31.27 (28.793)
  Diarrhea Score; Cycle 9 Day 1: number analyzed (Participants) | 91 | 92
  Diarrhea Score; Cycle 9 Day 1 | 34.43 (33.129) | 28.62 (28.637)
  Diarrhea Score; Cycle 10 Day 1: number analyzed (Participants) | 81 | 75
  Diarrhea Score; Cycle 10 Day 1 | 29.22 (29.992) | 29.33 (25.088)
  Diarrhea Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 72
  Diarrhea Score; Cycle 11 Day 1 | 28.02 (28.367) | 26.85 (26.619)
  Diarrhea Score; Cycle 12 Day 1: number analyzed (Participants) | 62 | 60
  Diarrhea Score; Cycle 12 Day 1 | 28.49 (31.273) | 22.78 (23.363)
  Diarrhea Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  Diarrhea Score; Cycle 13 Day 1 | 26.19 (28.223) | 23.03 (25.558)
  Diarrhea Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 52
  Diarrhea Score; Cycle 14 Day 1 | 26.53 (25.440) | 24.36 (22.008)
  Diarrhea Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 51
  Diarrhea Score; Cycle 15 Day 1 | 29.55 (29.828) | 30.07 (26.038)
  Diarrhea Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 47
  Diarrhea Score; Cycle 16 Day 1 | 20.33 (27.767) | 23.40 (21.886)
  Diarrhea Score; Cycle 17 Day 1: number analyzed (Participants) | 36 | 40
  Diarrhea Score; Cycle 17 Day 1 | 21.30 (24.107) | 29.17 (28.432)
  Diarrhea Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Diarrhea Score; Cycle 18 Day 1 | 21.51 (25.164) | 25.49 (23.296)
  Diarrhea Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Diarrhea Score; Cycle 19 Day 1 | 23.46 (28.963) | 21.57 (21.528)
  Diarrhea Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Diarrhea Score; Cycle 20 Day 1 | 19.75 (23.130) | 22.58 (23.392)
  Diarrhea Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Diarrhea Score; Cycle 21 Day 1 | 20.51 (26.795) | 21.43 (18.624)
  Diarrhea Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Diarrhea Score; Cycle 22 Day 1 | 17.54 (20.393) | 24.69 (19.812)
  Diarrhea Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Diarrhea Score; Cycle 23 Day 1 | 15.56 (17.213) | 22.22 (16.051)
  Diarrhea Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Diarrhea Score; Cycle 24 Day 1 | 11.11 (16.265) | 19.30 (16.909)
  Diarrhea Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Diarrhea Score; Cycle 25 Day 1 | 19.44 (22.285) | 18.75 (17.078)
  Diarrhea Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Diarrhea Score; Cycle 26 Day 1 | 25.00 (29.547) | 17.95 (17.296)
  Diarrhea Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Diarrhea Score; Cycle 27 Day 1 | 33.33 (21.082) | 33.33 (19.245)
  Diarrhea Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Diarrhea Score; Cycle 28 Day 1 | 16.67 (19.245) | 22.22 (17.213)
  Diarrhea Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Diarrhea Score; Cycle 29 Day 1 | 8.33 (16.667) | 20.00 (18.257)
  Diarrhea Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Diarrhea Score; Cycle 30 Day 1 | 16.67 (19.245) | 0
  Diarrhea Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Diarrhea Score; Cycle 31 Day 1 | 33.33 |
  Diarrhea Score; Off-treatment Visit: number analyzed (Participants) | 80 | 74
  Diarrhea Score; Off-treatment Visit | 18.33 (25.380) | 12.16 (19.565)
  Financial Difficulties Score; Baseline: number analyzed (Participants) | 170 | 162
  Financial Difficulties Score; Baseline | 21.76 (28.382) | 20.37 (29.076)
  Financial Difficulties Score; Cycle 2 Day 1: number analyzed (Participants) | 155 | 151
  Financial Difficulties Score; Cycle 2 Day 1 | 21.08 (28.177) | 15.01 (24.852)
  Financial Difficulties Score; Cycle 3 Day 1: number analyzed (Participants) | 147 | 141
  Financial Difficulties Score; Cycle 3 Day 1 | 23.13 (27.201) | 18.20 (27.451)
  Financial Difficulties Score; Cycle 4 Day 1: number analyzed (Participants) | 131 | 134
  Financial Difficulties Score; Cycle 4 Day 1 | 22.90 (27.761) | 16.42 (25.113)
  Financial Difficulties Score; Cycle 5 Day 1: number analyzed (Participants) | 125 | 126
  Financial Difficulties Score; Cycle 5 Day 1 | 22.93 (28.213) | 18.78 (29.058)
  Financial Difficulties Score; Cycle 6 Day 1: number analyzed (Participants) | 120 | 118
  Financial Difficulties Score; Cycle 6 Day 1 | 25.00 (27.416) | 17.80 (25.666)
  Financial Difficulties Score; Cycle 7 Day 1: number analyzed (Participants) | 105 | 105
  Financial Difficulties Score; Cycle 7 Day 1 | 30.16 (31.866) | 15.87 (24.062)
  Financial Difficulties Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 97
  Financial Difficulties Score; Cycle 8 Day 1 | 25.43 (29.176) | 17.53 (24.576)
  Financial Difficulties Score; Cycle 9 Day 1: number analyzed (Participants) | 90 | 90
  Financial Difficulties Score; Cycle 9 Day 1 | 25.56 (30.002) | 16.67 (23.440)
  Financial Difficulties Score; Cycle 10 Day 1: number analyzed (Participants) | 80 | 73
  Financial Difficulties Score; Cycle 10 Day 1 | 22.50 (27.952) | 17.35 (24.913)
  Financial Difficulties Score; Cycle 11 Day 1: number analyzed (Participants) | 66 | 72
  Financial Difficulties Score; Cycle 11 Day 1 | 26.26 (30.108) | 16.20 (24.382)
  Financial Difficulties Score; Cycle 12 Day 1: number analyzed (Participants) | 63 | 60
  Financial Difficulties Score; Cycle 12 Day 1 | 24.87 (28.061) | 16.11 (24.156)
  Financial Difficulties Score; Cycle 13 Day 1: number analyzed (Participants) | 55 | 54
  Financial Difficulties Score; Cycle 13 Day 1 | 23.03 (26.351) | 19.14 (25.577)
  Financial Difficulties Score; Cycle 14 Day 1: number analyzed (Participants) | 48 | 52
  Financial Difficulties Score; Cycle 14 Day 1 | 20.83 (22.413) | 17.31 (25.127)
  Financial Difficulties Score; Cycle 15 Day 1: number analyzed (Participants) | 43 | 51
  Financial Difficulties Score; Cycle 15 Day 1 | 21.71 (27.103) | 19.61 (26.813)
  Financial Difficulties Score; Cycle 16 Day 1: number analyzed (Participants) | 40 | 47
  Financial Difficulties Score; Cycle 16 Day 1 | 21.67 (25.654) | 17.02 (24.937)
  Financial Difficulties Score; Cycle 17 Day 1: number analyzed (Participants) | 35 | 40
  Financial Difficulties Score; Cycle 17 Day 1 | 23.81 (27.501) | 19.17 (27.099)
  Financial Difficulties Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 34
  Financial Difficulties Score; Cycle 18 Day 1 | 17.20 (18.995) | 19.61 (28.566)
  Financial Difficulties Score; Cycle 19 Day 1: number analyzed (Participants) | 27 | 34
  Financial Difficulties Score; Cycle 19 Day 1 | 18.52 (19.245) | 20.59 (28.444)
  Financial Difficulties Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 31
  Financial Difficulties Score; Cycle 20 Day 1 | 16.05 (21.424) | 20.43 (30.644)
  Financial Difficulties Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  Financial Difficulties Score; Cycle 21 Day 1 | 19.23 (21.444) | 20.24 (27.725)
  Financial Difficulties Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  Financial Difficulties Score; Cycle 22 Day 1 | 24.56 (24.450) | 20.99 (29.451)
  Financial Difficulties Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  Financial Difficulties Score; Cycle 23 Day 1 | 17.78 (17.213) | 23.61 (31.819)
  Financial Difficulties Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  Financial Difficulties Score; Cycle 24 Day 1 | 17.78 (21.331) | 19.30 (25.618)
  Financial Difficulties Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  Financial Difficulties Score; Cycle 25 Day 1 | 16.67 (22.473) | 16.67 (24.343)
  Financial Difficulties Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  Financial Difficulties Score; Cycle 26 Day 1 | 20.83 (24.801) | 20.51 (32.026)
  Financial Difficulties Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  Financial Difficulties Score; Cycle 27 Day 1 | 16.67 (18.257) | 0 (0)
  Financial Difficulties Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  Financial Difficulties Score; Cycle 28 Day 1 | 25.00 (16.667) | 0 (0)
  Financial Difficulties Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  Financial Difficulties Score; Cycle 29 Day 1 | 25.00 (16.667) | 0 (0)
  Financial Difficulties Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  Financial Difficulties Score; Cycle 30 Day 1 | 25.00 (16.667) | 0
  Financial Difficulties Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  Financial Difficulties Score; Cycle 31 Day 1 | 0 |
  Financial Difficulties Score; Off-treatment Visit: number analyzed (Participants) | 79 | 73
  Financial Difficulties Score; Off-treatment Visit | 31.65 (32.423) | 25.11 (30.318)

17. Secondary Outcome: HRQoL Assessed by European Quality of Life (EuroQol) Five-Dimensional, 3-Level (EQ-5D-3L) Index Score and Visual Analogue Scale (VAS)
Description: The EQ-5D-3L is a health profile questionnaire assessing quality of life along 5 dimensions. Participants rate 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 5-15 with "5" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. The EQ-5D index was calculated by applying preference-based weights (tariffs) to the scores of the five health state dimensions. Index values can range from -1 to 1, with 0 representing a health state equivalent to death and 1 representing perfect health. EQ-5D-3L also included an EQ visual analogue scale (VAS) that ranges between 100 (best imaginable health) and 0 (worst imaginable health). Decrease from baseline in EQ-5D-3L signifies improvement. Total index EQ-5D-3L summary score was weighted with a range of -0.594 (worst) to 1.0 (best).
Time Frame: as for outcome 15
Population: QoL analysis set consisted of all participants who had any QoL data. Here "overall number of participants analyzed" are the participants who were evaluable for the outcome measure and "number analyzed" were the participants who were evaluable at given time points. . As pre-specified in protocol, data for this secondary outcome measure was collected and analyzed till primary analysis only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 168 | 161
score on a scale
  EQ-5D Index Score; Baseline | 0.76 (0.216) | 0.78 (0.232)
  EQ-5D Index Score; Cycle 2 Day 1: number analyzed (Participants) | 151 | 147
  EQ-5D Index Score; Cycle 2 Day 1 | 0.76 (0.178) | 0.76 (0.230)
  EQ-5D Index Score; Cycle 3 Day 1: number analyzed (Participants) | 144 | 134
  EQ-5D Index Score; Cycle 3 Day 1 | 0.73 (0.232) | 0.78 (0.239)
  EQ-5D Index Score; Cycle 4 Day 1: number analyzed (Participants) | 131 | 131
  EQ-5D Index Score; Cycle 4 Day 1 | 0.73 (0.213) | 0.78 (0.236)
  EQ-5D Index Score; Cycle 5 Day 1: number analyzed (Participants) | 124 | 124
  EQ-5D Index Score; Cycle 5 Day 1 | 0.73 (0.212) | 0.78 (0.199)
  EQ-5D Index Score; Cycle 6 Day 1: number analyzed (Participants) | 121 | 114
  EQ-5D Index Score; Cycle 6 Day 1 | 0.73 (0.220) | 0.77 (0.225)
  EQ-5D Index Score; Cycle 7 Day 1: number analyzed (Participants) | 103 | 102
  EQ-5D Index Score; Cycle 7 Day 1 | 0.71 (0.219) | 0.78 (0.196)
  EQ-5D Index Score; Cycle 8 Day 1: number analyzed (Participants) | 95 | 95
  EQ-5D Index Score; Cycle 8 Day 1 | 0.75 (0.187) | 0.80 (0.187)
  EQ-5D Index Score; Cycle 9 Day 1: number analyzed (Participants) | 87 | 89
  EQ-5D Index Score; Cycle 9 Day 1 | 0.73 (0.192) | 0.79 (0.192)
  EQ-5D Index Score; Cycle 10 Day 1: number analyzed (Participants) | 77 | 71
  EQ-5D Index Score; Cycle 10 Day 1 | 0.76 (0.186) | 0.81 (0.177)
  EQ-5D Index Score; Cycle 11 Day 1: number analyzed (Participants) | 67 | 70
  EQ-5D Index Score; Cycle 11 Day 1 | 0.77 (0.185) | 0.82 (0.82)
  EQ-5D Index Score; Cycle 12 Day 1: number analyzed (Participants) | 64 | 59
  EQ-5D Index Score; Cycle 12 Day 1 | 0.77 (0.173) | 0.83 (0.161)
  EQ-5D Index Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 54
  EQ-5D Index Score; Cycle 13 Day 1 | 0.76 (0.157) | 0.82 (0.179)
  EQ-5D Index Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 51
  EQ-5D Index Score; Cycle 14 Day 1 | 0.77 (0.186) | 0.83 (0.163)
  EQ-5D Index Score; Cycle 15 Day 1: number analyzed (Participants) | 43 | 49
  EQ-5D Index Score; Cycle 15 Day 1 | 0.76 (0.191) | 0.81 (0.165)
  EQ-5D Index Score; Cycle 16 Day 1: number analyzed (Participants) | 40 | 46
  EQ-5D Index Score; Cycle 16 Day 1 | 0.73 (0.179) | 0.81 (0.212)
  EQ-5D Index Score; Cycle 17 Day 1: number analyzed (Participants) | 37 | 39
  EQ-5D Index Score; Cycle 17 Day 1 | 0.73 (0.211) | 0.83 (0.158)
  EQ-5D Index Score; Cycle 18 Day 1: number analyzed (Participants) | 31 | 33
  EQ-5D Index Score; Cycle 18 Day 1 | 0.76 (0.148) | 0.84 (0.177)
  EQ-5D Index Score; Cycle 19 Day 1: number analyzed (Participants) | 26 | 33
  EQ-5D Index Score; Cycle 19 Day 1 | 0.69 (0.266) | 0.79 (0.205)
  EQ-5D Index Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 30
  EQ-5D Index Score; Cycle 20 Day 1 | 0.70 (0.259) | 0.82 (0.167)
  EQ-5D Index Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  EQ-5D Index Score; Cycle 21 Day 1 | 0.73 (0.223) | 0.83 (0.180)
  EQ-5D Index Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  EQ-5D Index Score; Cycle 22 Day 1 | 0.74 (0.157) | 0.85 (0.173)
  EQ-5D Index Score; Cycle 23 Day 1: number analyzed (Participants) | 14 | 24
  EQ-5D Index Score; Cycle 23 Day 1 | 0.74 (0.149) | 0.82 (0.242)
  EQ-5D Index Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 18
  EQ-5D Index Score; Cycle 24 Day 1 | 0.75 (0.172) | 0.84 (0.156)
  EQ-5D Index Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  EQ-5D Index Score; Cycle 25 Day 1 | 0.70 (0.245) | 0.83 (0.175)
  EQ-5D Index Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  EQ-5D Index Score; Cycle 26 Day 1 | 0.72 (0.170) | 0.73 (0.438)
  EQ-5D Index Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 6
  EQ-5D Index Score; Cycle 27 Day 1 | 0.77 (0.135) | 0.93 (0.117)
  EQ-5D Index Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 5
  EQ-5D Index Score; Cycle 28 Day 1 | 0.73 (0.112) | 0.97 (0.067)
  EQ-5D Index Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 4
  EQ-5D Index Score; Cycle 29 Day 1 | 0.74 (0.120) | 0.96 (0.075)
  EQ-5D Index Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  EQ-5D Index Score; Cycle 30 Day 1 | 0.61 (0.391) | 1
  EQ-5D Index Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  EQ-5D Index Score; Cycle 31 Day 1 | 0.87 |
  EQ-5D Index Score; Off-treatment Visit: number analyzed (Participants) | 77 | 72
  EQ-5D Index Score; Off-treatment Visit | 0.61 (0.331) | 0.68 (0.314)
  EQ-VAS Score; Baseline: number analyzed (Participants) | 167 | 161
  EQ-VAS Score; Baseline | 68.57 (18.348) | 70.01 (20.552)
  EQ-VAS Score; Cycle 2 Day 1: number analyzed (Participants) | 149 | 147
  EQ-VAS Score; Cycle 2 Day 1 | 66.05 (18.531) | 69.52 (19.155)
  EQ-VAS Score; Cycle 3 Day 1: number analyzed (Participants) | 145 | 137
  EQ-VAS Score; Cycle 3 Day 1 | 66.22 (17.804) | 70.71 (17.648)
  EQ-VAS Score; Cycle 4 Day 1: number analyzed (Participants) | 130 | 133
  EQ-VAS Score; Cycle 4 Day 1 | 65.69 (18.265) | 69.66 (17.784)
  EQ-VAS Score; Cycle 5 Day 1: number analyzed (Participants) | 122 | 125
  EQ-VAS Score; Cycle 5 Day 1 | 65.86 (18.908) | 70.30 (19.492)
  EQ-VAS Score; Cycle 6 Day 1: number analyzed (Participants) | 118 | 116
  EQ-VAS Score; Cycle 6 Day 1 | 65.53 (20.027) | 71.73 (17.366)
  EQ-VAS Score; Cycle 7 Day 1: number analyzed (Participants) | 102 | 104
  EQ-VAS Score; Cycle 7 Day 1 | 65.74 (18.063) | 70.39 (19.387)
  EQ-VAS Score; Cycle 8 Day 1: number analyzed (Participants) | 97 | 95
  EQ-VAS Score; Cycle 8 Day 1 | 64.16 (18.969) | 70.40 (20.130)
  EQ-VAS Score; Cycle 9 Day 1: number analyzed (Participants) | 90 | 90
  EQ-VAS Score; Cycle 9 Day 1 | 65.51 (17.670) | 69.92 (19.452)
  EQ-VAS Score; Cycle 10 Day 1: number analyzed (Participants) | 77 | 73
  EQ-VAS Score; Cycle 10 Day 1 | 66.92 (17.747) | 73.18 (20.167)
  EQ-VAS Score; Cycle 11 Day 1: number analyzed (Participants) | 69 | 71
  EQ-VAS Score; Cycle 11 Day 1 | 67.74 (16.850) | 73.21 (19.310)
  EQ-VAS Score; Cycle 12 Day 1: number analyzed (Participants) | 65 | 61
  EQ-VAS Score; Cycle 12 Day 1 | 66.46 (18.680) | 74.46 (17.139)
  EQ-VAS Score; Cycle 13 Day 1: number analyzed (Participants) | 56 | 55
  EQ-VAS Score; Cycle 13 Day 1 | 65.64 (19.690) | 74.35 (17.766)
  EQ-VAS Score; Cycle 14 Day 1: number analyzed (Participants) | 49 | 53
  EQ-VAS Score; Cycle 14 Day 1 | 66.41 (17.839) | 74.40 (17.678)
  EQ-VAS Score; Cycle 15 Day 1: number analyzed (Participants) | 44 | 50
  EQ-VAS Score; Cycle 15 Day 1 | 67.05 (17.847) | 72.58 (19.060)
  EQ-VAS Score; Cycle 16 Day 1: number analyzed (Participants) | 41 | 46
  EQ-VAS Score; Cycle 16 Day 1 | 66.54 (18.118) | 72.80 (17.733)
  EQ-VAS Score; Cycle 17 Day 1: number analyzed (Participants) | 37 | 40
  EQ-VAS Score; Cycle 17 Day 1 | 65.78 (17.755) | 73.80 (17.593)
  EQ-VAS Score; Cycle 18 Day 1: number analyzed (Participants) | 30 | 34
  EQ-VAS Score; Cycle 18 Day 1 | 64.70 (18.170) | 73.71 (16.665)
  EQ-VAS Score; Cycle 19 Day 1: number analyzed (Participants) | 26 | 34
  EQ-VAS Score; Cycle 19 Day 1 | 62.15 (20.676) | 71.76 (19.272)
  EQ-VAS Score; Cycle 20 Day 1: number analyzed (Participants) | 27 | 30
  EQ-VAS Score; Cycle 20 Day 1 | 62.70 (19.779) | 72.07 (19.293)
  EQ-VAS Score; Cycle 21 Day 1: number analyzed (Participants) | 26 | 28
  EQ-VAS Score; Cycle 21 Day 1 | 62.12 (17.974) | 76.46 (16.836)
  EQ-VAS Score; Cycle 22 Day 1: number analyzed (Participants) | 19 | 27
  EQ-VAS Score; Cycle 22 Day 1 | 65.21 (14.722) | 74.44 (16.860)
  EQ-VAS Score; Cycle 23 Day 1: number analyzed (Participants) | 15 | 24
  EQ-VAS Score; Cycle 23 Day 1 | 67.73 (15.650) | 73.67 (17.704)
  EQ-VAS Score; Cycle 24 Day 1: number analyzed (Participants) | 15 | 19
  EQ-VAS Score; Cycle 24 Day 1 | 65.27 (19.381) | 71.21 (21.212)
  EQ-VAS Score; Cycle 25 Day 1: number analyzed (Participants) | 12 | 16
  EQ-VAS Score; Cycle 25 Day 1 | 60.58 (19.313) | 72.81 (16.897)
  EQ-VAS Score; Cycle 26 Day 1: number analyzed (Participants) | 8 | 13
  EQ-VAS Score; Cycle 26 Day 1 | 64.13 (16.313) | 65.23 (25.652)
  EQ-VAS Score; Cycle 27 Day 1: number analyzed (Participants) | 6 | 7
  EQ-VAS Score; Cycle 27 Day 1 | 61.83 (18.357) | 77.43 (16.762)
  EQ-VAS Score; Cycle 28 Day 1: number analyzed (Participants) | 4 | 6
  EQ-VAS Score; Cycle 28 Day 1 | 54.25 (8.694) | 77.50 (20.907)
  EQ-VAS Score; Cycle 29 Day 1: number analyzed (Participants) | 4 | 5
  EQ-VAS Score; Cycle 29 Day 1 | 52.75 (12.093) | 74 (21.036)
  EQ-VAS Score; Cycle 30 Day 1: number analyzed (Participants) | 4 | 1
  EQ-VAS Score; Cycle 30 Day 1 | 51.75 (11.295) | 50
  EQ-VAS Score; Cycle 31 Day 1: number analyzed (Participants) | 1 | 0
  EQ-VAS Score; Cycle 31 Day 1 | 35 |
  EQ-VAS Score; Off-treatment Visit: number analyzed (Participants) | 77 | 73
  EQ-VAS Score; Off-treatment Visit | 58.48 (23.516) | 62.66 (22.252)

18. Secondary Outcome: Progression-free Survival After Next Line of Therapy (PFS2)
Description: PFS2, defined as the time from randomization to the date of PD after next line of therapy or death from any cause, whichever occurred first based on investigator assessment according to RECIST v1.1. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. Median PFS2 was analyzed using the Kaplan-Meier product-limit estimates for each treatment group and presented with 2-sided 95% CI. As pre-specified in protocol, data for this secondary outcome measure was collected and analyzed till the primary analysis only.
Time Frame: From the time of randomization to the date of PD after next line of therapy or death from any cause or the date of data cutoff for the primary analysis, whichever occurs first (up to 29 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 156 | 155
months | 18.2 [13.1 to 22.5] | 19.5 [14.1 to 23.8]

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug up to 28 days after last dose of study drug (up to 71 months)
Description: Reported deaths included all anticipated and unanticipated deaths due to any cause in the study.
Groups:
- Lenvatinib 14 mg + Everolimus 5 mg: Participants received lenvatinib 14 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily as the starting dose for in a 28-day treatment cycle until progressive disease (PD), development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first. If there were no intolerable Grade 2 or any >= Grade 3 TEAEs that required dose reduction in the first 28-day cycle (that is, the first 4 weeks of treatment), lenvatinib dose was escalated to 18 mg once daily (along with everolimus 5 mg) beginning in Cycle 2 or later (cycle length = 28 days) during randomization phase.
- Lenvatinib 18 mg + Everolimus 5 mg: Participants received lenvatinib 18 mg, capsule, orally, once daily along with everolimus 5 mg, tablet, orally, once daily as the starting dose for in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first.
Arm/Group | Lenvatinib 14 mg + Everolimus 5 mg | Lenvatinib 18 mg + Everolimus 5 mg
All-Cause Mortality (participants affected / at risk) | 71/173 | 60/168
Serious Adverse Events (participants affected / at risk) | 92/173 | 87/168
Other Adverse Events (participants affected / at risk) | 172/173 | 166/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 14 mg + Everolimus 5 mg (N=173) | Lenvatinib 18 mg + Everolimus 5 mg (N=168)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (3)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (3) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 6 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9) | 2 (3)
Asthenia (General disorders) | 2 (3) | 2 (2)
Chest pain (General disorders) | 1 (2) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (2) | 2 (2)
Localised oedema (General disorders) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (4) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Malignant biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Paracancerous pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 13 (17) | 7 (9)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 3 (5) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 4 (5)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 5 (5)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 6 (10)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 14 mg + Everolimus 5 mg (N=173) | Lenvatinib 18 mg + Everolimus 5 mg (N=168)
Anaemia (Blood and lymphatic system disorders) | 37 (56) | 29 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (13) | 10 (29)
Hyperthyroidism (Endocrine disorders) | 5 (6) | 9 (11)
Hypothyroidism (Endocrine disorders) | 30 (38) | 35 (42)
Abdominal pain (Gastrointestinal disorders) | 29 (46) | 28 (40)
Abdominal pain upper (Gastrointestinal disorders) | 15 (20) | 13 (21)
Constipation (Gastrointestinal disorders) | 22 (25) | 25 (32)
Diarrhoea (Gastrointestinal disorders) | 117 (352) | 123 (394)
Dyspepsia (Gastrointestinal disorders) | 14 (21) | 15 (23)
Nausea (Gastrointestinal disorders) | 54 (104) | 52 (103)
Stomatitis (Gastrointestinal disorders) | 61 (120) | 49 (92)
Toothache (Gastrointestinal disorders) | 8 (10) | 11 (11)
Vomiting (Gastrointestinal disorders) | 41 (85) | 43 (85)
Asthenia (General disorders) | 42 (104) | 39 (100)
Fatigue (General disorders) | 51 (93) | 50 (104)
Oedema peripheral (General disorders) | 21 (31) | 23 (44)
Pyrexia (General disorders) | 17 (22) | 16 (21)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (12)
Urinary tract infection (Infections and infestations) | 11 (16) | 9 (14)
Alanine aminotransferase increased (Investigations) | 11 (21) | 14 (21)
Amylase increased (Investigations) | 9 (15) | 8 (12)
Aspartate aminotransferase increased (Investigations) | 13 (17) | 12 (16)
Blood alkaline phosphatase increased (Investigations) | 11 (11) | 9 (12)
Blood cholesterol increased (Investigations) | 13 (19) | 22 (37)
Blood creatinine increased (Investigations) | 23 (30) | 25 (42)
Blood thyroid stimulating hormone increased (Investigations) | 11 (17) | 5 (6)
Blood triglycerides increased (Investigations) | 7 (19) | 13 (36)
Lipase increased (Investigations) | 18 (33) | 16 (26)
Platelet count decreased (Investigations) | 9 (22) | 12 (20)
Weight decreased (Investigations) | 36 (63) | 41 (73)
Decreased appetite (Metabolism and nutrition disorders) | 64 (130) | 57 (137)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 31 (64) | 26 (49)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (20) | 12 (36)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 37 (112) | 38 (136)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (10) | 10 (18)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (11) | 13 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12) | 19 (31)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (11) | 11 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (18) | 13 (26)
Hypophosphataemia (Metabolism and nutrition disorders) | 16 (24) | 11 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (29) | 17 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (23) | 17 (26)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 12 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (20) | 5 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 13 (19)
Headache (Nervous system disorders) | 24 (34) | 20 (28)
Insomnia (Psychiatric disorders) | 12 (14) | 16 (19)
Proteinuria (Renal and urinary disorders) | 40 (133) | 66 (186)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 30 (47)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 24 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (23) | 25 (33)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 (36) | 24 (28)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24 (36) | 26 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 28 (41) | 29 (43)
Hypertension (Vascular disorders) | 54 (113) | 59 (101)
Hypotension (Vascular disorders) | 7 (7) | 10 (16)
Pneumonia (Infections and infestations) | 9 (9) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 9 (12) | 5 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (14) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03173560/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03173560/SAP_001.pdf